CLINICAL TRIAL: NCT01031069
Title: Safety and Immunogenicity of Cervarix™ in Human Immunodeficiency Virus Infected Females
Brief Title: Evaluation of Safety and Immunogenicity of a Human Papillomavirus (HPV) Vaccine in Human Immunodeficiency Virus (HIV) Infected Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 109823; 2013-003429-28 (EudraCT Number)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: Cervarix; Gardasil; Immunogenicity; Cervical cancer; Safety; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No

ARMS (4):
- HIV+/Cervarix Group (Experimental): HIV seropositive female subjects, between and including 15 and 25 years of age, who received 3 doses of Cervarix vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm, according to a three-dose schedule: at Day 0, Week 6, Month 6.
  Interventions: Biological: GSK Biologicals' HPV vaccine 580299
- HIV+/Gardasil Group (Active Comparator): HIV seropositive female subjects, between and including 15 and 25 years of age, who received 3 doses of Gardasil vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm, according to a three-dose schedule: at Day 0, Week 6, Month 6.
  Interventions: Biological: Merck's Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine (Gardasil)
- HIV-/Cervarix Group (Experimental): HIV seronegative female subjects, between and including 15 and 25 years of age, who received 3 doses of Cervarix vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm, according to a three-dose schedule: at Day 0, Week 6, Month 6.
  Interventions: Biological: GSK Biologicals' HPV vaccine 580299
- HIV-/Gardasil Group (Active Comparator): HIV seronegative female subjects, between and including 15 and 25 years of age, who received 3 doses of Gardasil vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm, according to a three-dose schedule: at Day 0, Week 6, Month 6.
  Interventions: Biological: Merck's Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine (Gardasil)

INTERVENTIONS:
Biological: GSK Biologicals' HPV vaccine 580299 — Subjects received three doses of the study vaccine administered intramuscularly according to a Day 0, Week 6, and Month 6 vaccination schedule.
  Other Names: Cervarix
  Arms: HIV+/Cervarix Group; HIV-/Cervarix Group
Biological: Merck's Human Papillomavirus Quadrivalent (Types 6, 11, 16, and 18) Vaccine (Gardasil) — Subjects received three doses of the study vaccine administered intramuscularly according to a Day 0, Week 6, and Month 6 vaccination schedule.
  Other Names: Gardasil
  Arms: HIV+/Gardasil Group; HIV-/Gardasil Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. This Phase IV, observer-blind study is designed to evaluate the safety and immunogenicity of Cervarix in HIV infected females aged 15 to 25 years as compared to Merck's HPV vaccine (Gardasil). For comparative purposes, a group of HIV negative females will also be evaluated. All subjects will receive the HPV vaccine (either Cervarix or Gardasil) according to a three-dose schedule (Day 0, Week 6, Month 6).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s)/legally acceptable representative(s) (LAR) can and will comply with the requirements of the protocol.
* A female between, and including, 15 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject and/or from the subject's parent or LAR.
* Subjects willing to undergo HIV Voluntary Counseling and Testing (VCT) and willing to be informed of their HIV infection status.
* For HIV seropositive subjects:

  * Subjects must be HIV seropositive according to World Health Organization (WHO) case definition.
  * Subject must be asymptomatic (or only have persistent generalized lymphadenopathy).
  * Subjects should have a CD4 cell count > 350 cells/mm3.
  * If currently taking antiretrovirals (ARVs), subjects must be on compliant to triple therapy (highly active ART) and have undetectable viral load on two previous clinical visits within the six months prior to study entry.
* For HIV seronegative subjects:

  * Subjects confirmed as HIV seronegative at the screening visit.
* For non-virgin female subjects:

  * Subjects must have no history of abnormal cytology or CIN 1/2/3.
  * Subjects must have had no more than six life-time sexual partners prior to enrollment.
* Subjects must have no history of congenital malformations of the uterine cervix, or history of cauterization or surgical procedures involving damage to the transformation zone of the cervix or stenosis.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at screening and on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (Day 0 to Month 24).
* ART not compliant with the National Guidelines.
* Active tuberculosis (TB) visit (criteria mandatory only for HIV+ subjects).
* Current TB therapy.
* Hemoglobin < 8.0 g/dL at the screening visit.
* Creatinine > 1.5-fold the upper limit of normal (ULN) at the screening visit.
* Alanine aminotransferase (ALT) > 2.5-fold ULN at the screening visit.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period (Day 0 to Month 24).
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs (with the exception of ART) within six months prior to the first vaccine dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days (Days 0 - 29) before the first dose of study vaccine/control. Enrollment will be postponed until the subject is outside the specified window.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before or 30 days after (i.e., Days 0 - 29) any dose of study vaccine.
* Previous administration of components of the investigational vaccine.
* Cancer or autoimmune disease under treatment.
* Hypersensitivity to latex.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine/control.
* Acute disease and/or fever at the time of enrollment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory testing performed at the screening visit.
* History of any neurological disorders or seizures.
* Pregnant or breastfeeding female.
* A subject planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose (i.e., up to Month 8).
* Concurrently participating in another clinical study, at any time during the study period (Day 0 to Month 24), in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any medically diagnosed or suspected immunodeficient condition (other than HIV for HIV seropositive subjects), based on medical history, physical examination and/or laboratory tests results.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine/control or planned administration during the study period. Enrollment will be postponed until the subject is outside the specified window.
* Administration of trimethoprim/sulphamethoxazole within seven days before the first dose of study vaccine/control, or planned administration of trimethoprim/sulphamethoxazole within seven days after the first dose of study vaccine/control.
* Current drugs or alcohol abuse.
* Child in care.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 873 (Actual)
Dates: Start 2010-10-26 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Brazil (5):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Estonia (2):
  - GSK Investigational Site, Kohtla-Järve
  - GSK Investigational Site, Tallinn
- India (4):
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20391

REFERENCES:
- [Background] Folschweiller N, Teixeira J, Joshi S, Goldani LZ, Supparatpinyo K, Basu P, Chotpitayasunondh T, Chetchotisakd P, Ruxrungtham K, Roteli-Martins C, Grinsztejn B, Quintana SM, Kumarasamy N, Poongulali S, Kulkarni V, Lin L, Datta SK, Descamps D, Dodet M, Dubin G, Friel D, Hezareh M, Karkada N, Meric Camilleri D, Poncelet S, Salaun B, Tavares-da-Silva F, Thomas-Jooris F, Struyf F. Immunogenicity and safety of the AS04-HPV-16/18 and HPV-6/11/16/18 human papillomavirus vaccines in asymptomatic young women living with HIV aged 15-25 years: A phase IV randomized comparative study. EClinicalMedicine. 2020 May 25;23:100353. doi: 10.1016/j.eclinm.2020.100353. eCollection 2020 Jun. PMID 32639485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A number of 873 subjects were enrolled, out of which 173 subjects were excluded from all statistical analysis.
  154 subjects were not administered any vaccine dose (146 screen failures subjects and 8 subjects that did not participate from Visit 1).
Pre-assignment Details: Screening involved: checking of inclusion/exclusion criteria, demographic data, history and physical examination, AF B sputum test and/or chest X-ray, blood sampling for HIV testing and safety, urine pregnancy testing, birth control and HIV, STI, STD counselling, checking records for concomitant medication/vaccination, subject card distribution.
Period: Overall Study
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Started | 129 | 128 | 144 | 145
Completed | 117 | 117 | 103 | 111
Not Completed | 12 | 11 | 41 | 34
Not completed — Serious Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 18 | 18
Not completed — Migrated/moved from study area | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 9 | 5 | 21 | 15
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group | Total
Number analyzed (Participants) | 129 | 128 | 144 | 145 | 546
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.4 (3.4) | 20.1 (3.5) | 19.3 (3.0) | 19.6 (3.0) | 19.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 128 | 144 | 145 | 546
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 10 | 6 | 4 | 4 | 24
  Asian - Central/South Asian Heritage | 20 | 18 | 67 | 68 | 173
  Asian - East Asian Heritage | 3 | 2 | 1 | 0 | 6
  Asian - Japanese Heritage | 0 | 0 | 1 | 2 | 3
  Asian - South East Asian Heritage | 40 | 44 | 39 | 42 | 165
  White - Arabic/North African Heritage | 17 | 12 | 7 | 6 | 42
  White - Caucasian/European Heritage | 33 | 37 | 24 | 19 | 113
  Unspecified | 6 | 9 | 1 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Human Immunodeficiency Virus Positive Subjects (HIV+) With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness, swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling with a maximum diameter greater than 50 millimeters (mm).
Time Frame: During the 7-day follow-up period (from the day of vaccination up to 6 subsequent days) after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had available symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 128 | 127
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 128 | 125
  Any Pain, Dose 1 | 115 | 58
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Pain, Dose 1 | 4 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 128 | 125
  Any Redness, Dose 1 | 24 | 19
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 128 | 125
  Any Swelling, Dose 1 | 25 | 6
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Swelling, Dose 1 | 2 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 127 | 125
  Any Pain, Dose 2 | 98 | 56
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Pain, Dose 2 | 5 | 6
  Any Redness, Dose 2: number analyzed (Participants) | 127 | 125
  Any Redness, Dose 2 | 18 | 13
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 127 | 125
  Any Swelling, Dose 2 | 16 | 11
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 117 | 117
  Any Pain, Dose 3 | 87 | 60
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Pain, Dose 3 | 5 | 2
  Any Redness, Dose 3: number analyzed (Participants) | 117 | 117
  Any Redness, Dose 3 | 17 | 18
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Redness, Dose 3 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 117 | 117
  Any Swelling, Dose 3 | 19 | 10
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Swelling, Dose 3 | 1 | 0
  Any Pain, Across Doses | 120 | 85
  Grade 3 Pain, Across Doses | 11 | 6
  Any Redness, Across Doses | 41 | 34
  Grade 3 Redness, Across Doses | 1 | 0
  Any Swelling, Across Doses | 38 | 20
  Grade 3 Swelling, Across Doses | 2 | 0

2. Primary Outcome: Number of HIV+ Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal [nausea, vomiting, diarrhoea and/or abdominal pain], headache, myalgia, rash, temperature [defined as axillary temperature higher than (>) 37.5 degrees Celsius (°C)] and urticaria. Any = occurrence of the symptom regardless of intensity grade and relationship. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature > 39.0 °C. Grade 3 urticaria = urticaria distributed on at least 4 body areas. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 128 | 127
Participants
  Any Arthralgia, Dose 1: number analyzed (Participants) | 128 | 125
  Any Arthralgia, Dose 1 | 29 | 20
  Grade 3 Arthralgia, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Arthralgia, Dose 1 | 1 | 1
  Related Arthralgia, Dose 1: number analyzed (Participants) | 128 | 125
  Related Arthralgia, Dose 1 | 19 | 13
  Any Fatigue, Dose 1: number analyzed (Participants) | 128 | 125
  Any Fatigue, Dose 1 | 50 | 47
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Fatigue, Dose 1 | 4 | 0
  Related Fatigue, Dose 1: number analyzed (Participants) | 128 | 125
  Related Fatigue, Dose 1 | 30 | 29
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 128 | 125
  Any Gastrointestinal, Dose 1 | 30 | 21
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Gastrointestinal, Dose 1 | 2 | 0
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 128 | 125
  Related Gastrointestinal, Dose 1 | 19 | 15
  Any Headache, Dose 1: number analyzed (Participants) | 128 | 125
  Any Headache, Dose 1 | 61 | 48
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Headache, Dose 1 | 4 | 1
  Related Headache, Dose 1: number analyzed (Participants) | 128 | 125
  Related Headache, Dose 1 | 39 | 27
  Any Myalgia, Dose 1: number analyzed (Participants) | 128 | 125
  Any Myalgia, Dose 1 | 49 | 34
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Myalgia, Dose 1 | 2 | 1
  Related Myalgia, Dose 1: number analyzed (Participants) | 128 | 125
  Related Myalgia, Dose 1 | 35 | 25
  Any Rash, Dose 1: number analyzed (Participants) | 128 | 125
  Any Rash, Dose 1 | 7 | 4
  Grade 3 Rash, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Rash, Dose 1 | 1 | 0
  Related Rash, Dose 1: number analyzed (Participants) | 128 | 125
  Related Rash, Dose 1 | 4 | 0
  Any Temperature, Dose 1: number analyzed (Participants) | 128 | 125
  Any Temperature, Dose 1 | 9 | 5
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 128 | 125
  Related Temperature, Dose 1 | 7 | 4
  Any Urticaria, Dose 1: number analyzed (Participants) | 128 | 125
  Any Urticaria, Dose 1 | 8 | 3
  Grade 3 Urticaria, Dose 1: number analyzed (Participants) | 128 | 125
  Grade 3 Urticaria, Dose 1 | 0 | 0
  Related Urticaria, Dose 1: number analyzed (Participants) | 128 | 125
  Related Urticaria, Dose 1 | 6 | 3
  Any Arthralgia, Dose 2: number analyzed (Participants) | 127 | 125
  Any Arthralgia, Dose 2 | 18 | 21
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Arthralgia, Dose 2 | 0 | 3
  Related Arthralgia, Dose 2: number analyzed (Participants) | 127 | 125
  Related Arthralgia, Dose 2 | 11 | 14
  Any Fatigue, Dose 2: number analyzed (Participants) | 127 | 125
  Any Fatigue, Dose 2 | 38 | 40
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Fatigue, Dose 2 | 2 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 127 | 125
  Related Fatigue, Dose 2 | 20 | 25
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 127 | 125
  Any Gastrointestinal, Dose 2 | 15 | 17
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 127 | 125
  Related Gastrointestinal, Dose 2 | 11 | 11
  Any Headache, Dose 2: number analyzed (Participants) | 127 | 125
  Any Headache, Dose 2 | 48 | 37
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Headache, Dose 2 | 5 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 127 | 125
  Related Headache, Dose 2 | 30 | 20
  Any Myalgia, Dose 2: number analyzed (Participants) | 127 | 125
  Any Myalgia, Dose 2 | 36 | 26
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Myalgia, Dose 2 | 2 | 4
  Related Myalgia, Dose 2: number analyzed (Participants) | 127 | 125
  Related Myalgia, Dose 2 | 25 | 19
  Any Rash, Dose 2: number analyzed (Participants) | 127 | 125
  Any Rash, Dose 2 | 2 | 1
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Rash, Dose 2 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 127 | 125
  Related Rash, Dose 2 | 0 | 0
  Any Temperature, Dose 2: number analyzed (Participants) | 127 | 125
  Any Temperature, Dose 2 | 11 | 4
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 127 | 125
  Related Temperature, Dose 2 | 9 | 2
  Any Urticaria, Dose 2: number analyzed (Participants) | 127 | 125
  Any Urticaria, Dose 2 | 5 | 4
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 127 | 125
  Grade 3 Urticaria, Dose 2 | 1 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 127 | 125
  Related Urticaria, Dose 2 | 4 | 4
  Any Arthralgia, Dose 3: number analyzed (Participants) | 117 | 117
  Any Arthralgia, Dose 3 | 17 | 15
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Arthralgia, Dose 3 | 2 | 1
  Related Arthralgia, Dose 3: number analyzed (Participants) | 117 | 117
  Related Arthralgia, Dose 3 | 13 | 12
  Any Fatigue, Dose 3: number analyzed (Participants) | 117 | 117
  Any Fatigue, Dose 3 | 40 | 31
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Fatigue, Dose 3 | 1 | 1
  Related Fatigue, Dose 3: number analyzed (Participants) | 117 | 117
  Related Fatigue, Dose 3 | 30 | 22
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 117 | 117
  Any Gastrointestinal, Dose 3 | 13 | 17
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Gastrointestinal, Dose 3 | 1 | 1
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 117 | 117
  Related Gastrointestinal, Dose 3 | 9 | 13
  Any Headache, Dose 3: number analyzed (Participants) | 117 | 117
  Any Headache, Dose 3 | 48 | 27
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Headache, Dose 3 | 2 | 2
  Related Headache, Dose 3: number analyzed (Participants) | 117 | 117
  Related Headache, Dose 3 | 39 | 16
  Any Myalgia, Dose 3: number analyzed (Participants) | 117 | 117
  Any Myalgia, Dose 3 | 30 | 21
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Myalgia, Dose 3 | 4 | 1
  Related Myalgia, Dose 3: number analyzed (Participants) | 117 | 117
  Related Myalgia, Dose 3 | 26 | 17
  Any Rash, Dose 3: number analyzed (Participants) | 117 | 117
  Any Rash, Dose 3 | 2 | 1
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Rash, Dose 3 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 117 | 117
  Related Rash, Dose 3 | 1 | 0
  Any Temperature, Dose 3: number analyzed (Participants) | 117 | 117
  Any Temperature, Dose 3 | 10 | 12
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Temperature, Dose 3 | 1 | 1
  Related Temperature, Dose 3: number analyzed (Participants) | 117 | 117
  Related Temperature, Dose 3 | 7 | 6
  Any Urticaria, Dose 3: number analyzed (Participants) | 117 | 117
  Any Urticaria, Dose 3 | 2 | 4
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 117 | 117
  Grade 3 Urticaria, Dose 3 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 117 | 117
  Related Urticaria, Dose 3 | 2 | 2
  Any Arthralgia, Across Doses | 41 | 38
  Grade 3 Arthralgia, Across Doses | 3 | 4
  Related Arthralgia, Across Doses | 31 | 28
  Any Fatigue, Across Doses | 73 | 59
  Grade 3 Fatigue, Across Doses | 6 | 2
  Related Fatigue, Across Doses | 50 | 39
  Any Gastrointestinal, Across Doses | 41 | 35
  Grade 3 Gastrointestinal, Across Doses | 3 | 1
  Related Gastrointestinal, Across Doses | 27 | 23
  Any Headache, Across Doses | 88 | 63
  Grade 3 Headache, Across Doses | 11 | 4
  Related Headache, Across Doses | 65 | 39
  Any Myalgia, Across Doses | 68 | 51
  Grade 3 Myalgia, Across Doses | 7 | 4
  Related Myalgia, Across Doses | 52 | 37
  Any Rash, Across Doses | 11 | 5
  Grade 3 Rash, Across Doses | 1 | 0
  Related Rash, Across Doses | 5 | 0
  Any Temperature, Across Doses | 23 | 19
  Grade 3 Temperature, Across Doses | 1 | 1
  Related Temperature, Across Doses | 18 | 10
  Any Urticaria, Across Doses | 13 | 9
  Grade 3 Urticaria, Across Doses | 1 | 0
  Related Urticaria, Across Doses | 10 | 8

3. Primary Outcome: Number of HIV+ Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day follow-up period (from the day of vaccination up to 29 subsequent days) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort for analysis of safety, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants
  Any AE(s) | 41 | 41
  Grade 3 AE(s) | 7 | 4
  Related AE(s) | 9 | 8

4. Primary Outcome: Number of HIV+ Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or represented a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants | 6 | 6

5. Primary Outcome: Number of HIV+ Subjects With Medically Significant Conditions (MSCs)
Description: Medically significant conditions (MSCs) are defined as AEs prompting emergency room or physician visits that were not related to common diseases, or not related to routine visits for physical examination or vaccination, SAEs that were not related to common diseases.
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants | 17 | 27

6. Primary Outcome: Number of HIV+ Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants | 1 | 0

7. Primary Outcome: Number of HIV+ Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: Pregnancy related outcomes were: live infant no apparent congenital anomaly, live infant congenital anomaly, elective termination (termin.) no apparent congenital anomaly, elective termination (termin.) congenital anomaly, ectopic pregnancy, spontaneous abortion no apparent congenital (congen.) anomaly, stillbirth no apparent congenital anomaly, stillbirth congenital anomaly, lost to follow-up, pregnancy ongoing, missing.
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who reported any pregnancies and outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 4 | 2
Participants
  Live infant NO apparent congenital anomaly | 3 | 1
  Live infant congenital anomaly | 0 | 0
  Elective termin. NO apparent congenital anomaly | 0 | 0
  Elective termin. congenital anomaly | 0 | 0
  Ectopic pregnancy | 0 | 0
  Spontaneous abortion NO apparent congen. anomaly | 1 | 1
  Stillbirth NO apparent congenital anomaly | 0 | 0
  Stillbirth congenital anomaly | 0 | 0
  Lost to follow-up | 0 | 0
  Pregnancy ongoing | 0 | 0
  Missing | 0 | 0

8. Primary Outcome: Number of HIV+ Subjects With Haematological and Biochemical Parameter Abnormalities
Description: Among assessed haematological and biochemical parameters were: alanine aminotransferase [ALAT], basophilis [BSPH], creatinine [CRT], eosinophils [ESPH], haematocrit [HTCR], haemoglobin [HGB], lymphocytes [LYMP], monocytes [MONO], neutrophils [NTPH], platelets [PLAT], red blood cells [RBC] and white blood cells [WBC]. Unknown = value unknown for the specified visit and laboratory parameter; Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available at Month 7.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 121 | 121
Participants
  ALAT, Unknown | 0 | 0
  ALAT, Below | 4 | 3
  ALAT, Within | 110 | 105
  ALAT, Above | 7 | 13
  BSPH, Unknown | 0 | 0
  BSPH, Below | 0 | 0
  BSPH, Within | 120 | 121
  BSPH, Above | 1 | 0
  CRT, Unknown: number analyzed (Participants) | 121 | 120
  CRT, Unknown | 0 | 0
  CRT, Below: number analyzed (Participants) | 121 | 120
  CRT, Below | 29 | 36
  CRT, Within: number analyzed (Participants) | 121 | 120
  CRT, Within | 91 | 84
  CRT, Above: number analyzed (Participants) | 121 | 120
  CRT, Above | 1 | 0
  ESPH, Unknown | 0 | 0
  ESPH, Below | 9 | 10
  ESPH, Within | 108 | 106
  ESPH, Above | 4 | 5
  HTCR, Unknown | 0 | 0
  HTCR, Below | 19 | 27
  HTCR, Within | 101 | 92
  HTCR, Above | 1 | 2
  HGB, Unknown | 0 | 0
  HGB, Below | 28 | 37
  HGB, Within | 92 | 83
  HGB, Above | 1 | 1
  LYMP, Unknown | 0 | 0
  LYMP, Below | 12 | 11
  LYMP, Within | 96 | 97
  LYMP, Above | 13 | 13
  MONO, Unknown | 0 | 0
  MONO, Below | 4 | 7
  MONO, Within | 106 | 97
  MONO, Above | 11 | 17
  NTPH, Unknown | 0 | 0
  NTPH, Below | 16 | 17
  NTPH, Within | 97 | 93
  NTPH, Above | 8 | 11
  PLAT, Unknown | 0 | 0
  PLAT, Below | 1 | 3
  PLAT, Within | 118 | 114
  PLAT, Above | 2 | 4
  RBC, Unknown | 0 | 0
  RBC, Below | 36 | 34
  RBC, Within | 82 | 84
  RBC, Above | 3 | 3
  WBC, Unknown | 0 | 0
  WBC, Below | 10 | 9
  WBC, Within | 106 | 108
  WBC, Above | 5 | 4

9. Primary Outcome: Cluster of Differentiation 4 (CD4+) Cell Count in HIV+ Subjects at Month 7
Description: CD4+ cell count, expressed in cells/cubic millimeter (mm3), was assessed for HIV+ subjects.
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 121 | 121
cells/mm3 | 554.0 [440.0 to 799.0] | 568.0 [457.0 to 773.4]

10. Primary Outcome: HIV Viral Load (VL) in HIV+ Subjects at Month 7
Description: HIV VL, expressed in HIV copies/milliliter (mL), was assessed for HIV+ subjects.
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: HIV copies/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 96 | 95
HIV copies/mL | 1.9 [1.3 to 3.8] | 2.5 [1.3 to 3.8]

11. Primary Outcome: Number of HIV+ Subjects by World Health Organization (WHO) HIV Clinical Staging
Description: HIV+ subjects were categorised into clinical stages 1 through 4, as per the WHO classification [WHO, 2009].
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants
  Clinical Stage 1 | 113 | 114
  Clinical Stage 2 | 6 | 2
  Clinical Stage 3 | 1 | 1
  Clinical Stage 4 | 1 | 4

12. Primary Outcome: Pseudovirion-Based Neutralization Assay (PBNA) Titers of Anti-HPV-16/18 Antibodies in HIV+ Subjects, Based on Adapted According-to-protocol (ATP) Cohort for Immunogenicity
Description: Titers of anti-HPV-16/18 antibodies, expressed as Geometric Mean Titers (GMTs), with cut-offs greater than or equal to (≥) 40 estimated dose giving 50% signal reduction when compared to a control without serum (ED50), as assessed by the Pseudovirion-Based Neutralization Assay [PBNA], in HIV+ subjects.
  Between-group comparisons to assess non-inferiority were performed on the ATP cohort for immunogenicity (by PBNA, regardless of HPV serostatus at baseline).
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria and for whom Month 7 data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity at Month 7 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 79 | 83
Titers
  Anti-HPV-16 | 23436.1 [18186.4 to 30201.1] | 7507.0 [5378.1 to 10478.6]
  Anti-HPV-18: number analyzed (Participants) | 79 | 82
  Anti-HPV-18 | 12490.9 [9681.7 to 16115.2] | 1459.6 [965.4 to 2206.7]
Statistical Analysis 1: Comparison: HIV+/Cervarix Group vs HIV+/Gardasil Group; Adjusted GMT ratios for anti-HPV-16 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV+/Cervarix Group) was non-inferior to that of Gardasil vaccine (HIV+/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-16, measured by Pseudovirion-based neutralization assay (PBNA) one month after the administration of the third dose of vaccine in HIV+ subjects; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% confidence interval (CI) for the ratio of GMTs (Cervarix over Gardasil) being above (>) 0.5 for HPV-16 type; Adjusted GMT ratio = 2.95, 95% CI 2-sided [1.92 to 4.52]; Primary objectives were to be assessed sequentially: firstly, non-inferiority for both HPV-16 and HPV-18, and then, superiority for HPV-18 followed by superiority for HPV-16
Statistical Analysis 2: Comparison: HIV+/Cervarix Group vs HIV+/Gardasil Group; Adjusted GMT ratios for anti-HPV-18 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV+/Cervarix Group) was non-inferior to that of Gardasil vaccine (HIV+/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-18, measured by Pseudovirion-based neutralization assay (PBNA) one month after the administration of the third dose of vaccine in HIV+ subjects; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% confidence interval (CI) for the ratio of GMTs (Cervarix over Gardasil) being above (>) 0.5 for HPV-18 type; Adjusted GMT ratio = 7.83, 95% CI 2-sided [4.84 to 12.66]; [other analysis details as in outcome 12, analysis 1]

13. Primary Outcome: Pseudovirion-Based Neutralization Assay (PBNA) Titers of Anti-HPV-16/18 Antibodies in HIV+ Subjects, Based on Total Vaccinated Cohort (TVC)
Description: Titers of anti-HPV-16/18 antibodies, expressed as Geometric Mean Titers (GMTs), with cut-offs greater than or equal to (≥) 40 estimated dose giving 50% signal reduction when compared to a control without serum (ED50), as assessed by the Pseudovirion-Based Neutralization Assay [PBNA], in HIV+ subjects.
  Between-group comparisons to assess superiority were performed on the TVC (by PBNA, regardless of HPV serostatus at baseline).
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: The analysis was performed on the TVC for analysis of immunogenicity, which included vaccinated subjects for whom data concerning immunogenicity endpoint measures were available at Month 7.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 108 | 109
Titers
  Anti-HPV-16 | 21106.6 [15961.3 to 27910.6] | 7533.7 [5616.7 to 10105.0]
  Anti-HPV-18 | 11580.5 [8851.5 to 15150.9] | 1451.9 [1009.0 to 2089.2]
Statistical Analysis 1: Comparison: HIV+/Cervarix Group vs HIV+/Gardasil Group; Adjusted GMT ratios for anti-HPV-18 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV+/Cervarix Group) was superior to that of Gardasil vaccine (HIV+/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-18, measured by Pseudovirion-based neutralization assay (PBNA) in HIV+ subjects, assessed following a sequential approach; Test type: Superiority — Superiority was defined as the lower limit of the 95% CI for the ratio of GMTs (Cervarix over Gardasil) being above 1 for HPV-18 type, with a statistically significant p-value; p < 0.0001, ANOVA; ANOVA model on the log10 transformation of the titers for HIV+ subjects and including the vaccine group as fixed effect; Adjusted GMT ratio = 7.44, 95% CI 2-sided [4.79 to 11.54]; [other analysis details as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: HIV+/Cervarix Group vs HIV+/Gardasil Group; Adjusted GMT ratios for anti-HPV-16 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV+/Cervarix Group) was superior to that of Gardasil vaccine (HIV+/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-16, measured by Pseudovirion-based neutralization assay (PBNA) in HIV+ subjects, following a sequential approach; Test type: Superiority — Superiority was defined as the lower limit of the 95% CI for the ratio of GMTs (Cervarix over Gardasil) being above 1 for HPV-16 type, with a statistically significant p-value; p < 0.0001, ANOVA; ANOVA model on the log10 transformation of the titers for HIV+ subjects and including the vaccine group as fixed effect; Adjusted GMT ratio = 2.74, 95% CI 2-sided [1.83 to 4.11]; [other analysis details as in outcome 12, analysis 1]

14. Secondary Outcome: Number of HIV- Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 141 | 144
Participants
  Any Pain, Dose 1 | 127 | 91
  Grade 3 Pain, Dose 1 | 10 | 1
  Any Redness, Dose 1 | 32 | 21
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 23 | 14
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 136 | 139
  Any Pain, Dose 2 | 108 | 92
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Pain, Dose 2 | 6 | 2
  Any Redness, Dose 2: number analyzed (Participants) | 136 | 139
  Any Redness, Dose 2 | 29 | 29
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 136 | 139
  Any Swelling, Dose 2 | 24 | 27
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 125 | 129
  Any Pain, Dose 3 | 94 | 82
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Pain, Dose 3 | 10 | 6
  Any Redness, Dose 3: number analyzed (Participants) | 125 | 129
  Any Redness, Dose 3 | 28 | 19
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Redness, Dose 3 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 125 | 129
  Any Swelling, Dose 3 | 29 | 19
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across Doses | 133 | 119
  Grade 3 Pain, Across Doses | 22 | 8
  Any Redness, Across Doses | 52 | 42
  Grade 3 Redness, Across Doses | 0 | 0
  Any Swelling, Across Doses | 47 | 39
  Grade 3 Swelling, Across Doses | 0 | 0

15. Secondary Outcome: Number of HIV- Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 141 | 144
Participants
  Any Arthralgia, Dose 1 | 17 | 21
  Grade 3 Arthralgia, Dose 1 | 0 | 0
  Related Arthralgia, Dose 1 | 9 | 11
  Any Fatigue, Dose 1 | 45 | 34
  Grade 3 Fatigue, Dose 1 | 3 | 2
  Related Fatigue, Dose 1 | 29 | 17
  Any Gastrointestinal, Dose 1 | 19 | 14
  Grade 3 Gastrointestinal, Dose 1 | 1 | 1
  Related Gastrointestinal, Dose 1 | 8 | 11
  Any Headache, Dose 1 | 45 | 45
  Grade 3 Headache, Dose 1 | 0 | 2
  Related Headache, Dose 1 | 29 | 22
  Any Myalgia, Dose 1 | 44 | 36
  Grade 3 Myalgia, Dose 1 | 1 | 2
  Related Myalgia, Dose 1 | 28 | 21
  Any Rash, Dose 1 | 2 | 6
  Grade 3 Rash, Dose 1 | 0 | 0
  Related Rash, Dose 1 | 2 | 2
  Any Temperature, Dose 1 | 11 | 8
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 7 | 5
  Any Urticaria, Dose 1 | 3 | 3
  Grade 3 Urticaria, Dose 1 | 0 | 0
  Related Urticaria, Dose 1 | 3 | 3
  Any Arthralgia, Dose 2: number analyzed (Participants) | 136 | 139
  Any Arthralgia, Dose 2 | 14 | 12
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Arthralgia, Dose 2 | 0 | 0
  Related Arthralgia, Dose 2: number analyzed (Participants) | 136 | 139
  Related Arthralgia, Dose 2 | 9 | 5
  Any Fatigue, Dose 2: number analyzed (Participants) | 136 | 139
  Any Fatigue, Dose 2 | 34 | 34
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Fatigue, Dose 2 | 2 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 136 | 139
  Related Fatigue, Dose 2 | 19 | 19
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 136 | 139
  Any Gastrointestinal, Dose 2 | 9 | 15
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Gastrointestinal, Dose 2 | 1 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 136 | 139
  Related Gastrointestinal, Dose 2 | 7 | 6
  Any Headache, Dose 2: number analyzed (Participants) | 136 | 139
  Any Headache, Dose 2 | 35 | 31
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Headache, Dose 2 | 5 | 2
  Related Headache, Dose 2: number analyzed (Participants) | 136 | 139
  Related Headache, Dose 2 | 23 | 19
  Any Myalgia, Dose 2: number analyzed (Participants) | 136 | 139
  Any Myalgia, Dose 2 | 36 | 26
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Myalgia, Dose 2 | 1 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 136 | 139
  Related Myalgia, Dose 2 | 28 | 19
  Any Rash, Dose 2: number analyzed (Participants) | 136 | 139
  Any Rash, Dose 2 | 2 | 4
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Rash, Dose 2 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 136 | 139
  Related Rash, Dose 2 | 1 | 1
  Any Temperature, Dose 2: number analyzed (Participants) | 136 | 139
  Any Temperature, Dose 2 | 10 | 10
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Temperature, Dose 2 | 1 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 136 | 139
  Related Temperature, Dose 2 | 5 | 8
  Any Urticaria, Dose 2: number analyzed (Participants) | 136 | 139
  Any Urticaria, Dose 2 | 1 | 1
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 136 | 139
  Grade 3 Urticaria, Dose 2 | 0 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 136 | 139
  Related Urticaria, Dose 2 | 1 | 1
  Any Arthralgia, Dose 3: number analyzed (Participants) | 125 | 129
  Any Arthralgia, Dose 3 | 9 | 14
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Arthralgia, Dose 3 | 0 | 2
  Related Arthralgia, Dose 3: number analyzed (Participants) | 125 | 129
  Related Arthralgia, Dose 3 | 9 | 11
  Any Fatigue, Dose 3: number analyzed (Participants) | 125 | 129
  Any Fatigue, Dose 3 | 32 | 20
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Fatigue, Dose 3 | 1 | 2
  Related Fatigue, Dose 3: number analyzed (Participants) | 125 | 129
  Related Fatigue, Dose 3 | 29 | 15
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 125 | 129
  Any Gastrointestinal, Dose 3 | 7 | 9
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Gastrointestinal, Dose 3 | 1 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 125 | 129
  Related Gastrointestinal, Dose 3 | 6 | 6
  Any Headache, Dose 3: number analyzed (Participants) | 125 | 129
  Any Headache, Dose 3 | 33 | 25
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Headache, Dose 3 | 3 | 2
  Related Headache, Dose 3: number analyzed (Participants) | 125 | 129
  Related Headache, Dose 3 | 26 | 17
  Any Myalgia, Dose 3: number analyzed (Participants) | 125 | 129
  Any Myalgia, Dose 3 | 26 | 28
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Myalgia, Dose 3 | 2 | 2
  Related Myalgia, Dose 3: number analyzed (Participants) | 125 | 129
  Related Myalgia, Dose 3 | 22 | 21
  Any Rash, Dose 3: number analyzed (Participants) | 125 | 129
  Any Rash, Dose 3 | 2 | 0
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Rash, Dose 3 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 125 | 129
  Related Rash, Dose 3 | 2 | 0
  Any Temperature, Dose 3: number analyzed (Participants) | 125 | 129
  Any Temperature, Dose 3 | 9 | 10
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Temperature, Dose 3 | 2 | 1
  Related Temperature, Dose 3: number analyzed (Participants) | 125 | 129
  Related Temperature, Dose 3 | 7 | 6
  Any Urticaria, Dose 3: number analyzed (Participants) | 125 | 129
  Any Urticaria, Dose 3 | 2 | 3
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 125 | 129
  Grade 3 Urticaria, Dose 3 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 125 | 129
  Related Urticaria, Dose 3 | 2 | 3
  Any Arthralgia, Across Doses | 31 | 34
  Grade 3 Arthralgia, Across Doses | 0 | 2
  Related Arthralgia, Across Doses | 20 | 18
  Any Fatigue, Across Doses | 65 | 56
  Grade 3 Fatigue, Across Doses | 5 | 4
  Related Fatigue, Across Doses | 45 | 33
  Any Gastrointestinal, Across Doses | 28 | 26
  Grade 3 Gastrointestinal, Across Doses | 2 | 1
  Related Gastrointestinal, Across Doses | 17 | 17
  Any Headache, Across Doses | 69 | 67
  Grade 3 Headache, Across Doses | 7 | 5
  Related Headache, Across Doses | 51 | 40
  Any Myalgia, Across Doses | 64 | 53
  Grade 3 Myalgia, Across Doses | 3 | 4
  Related Myalgia, Across Doses | 44 | 40
  Any Rash, Across Doses | 5 | 8
  Grade 3 Rash, Across Doses | 0 | 0
  Related Rash, Across Doses | 5 | 3
  Any Temperature, Across Doses | 22 | 24
  Grade 3 Temperature, Across Doses | 3 | 1
  Related Temperature, Across Doses | 16 | 16
  Any Urticaria, Across Doses | 4 | 6
  Grade 3 Urticaria, Across Doses | 0 | 0
  Related Urticaria, Across Doses | 4 | 6

16. Secondary Outcome: Number of HIV- Subjects With Unsolicited Adverse Events (AEs)
Description: as for outcome 3
Time Frame: During the 30-day follow-up period (from the day of vaccination up to 29 subsequent days) after any vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 144 | 145
Participants
  Any AE(s) | 26 | 32
  Grade 3 AE(s) | 1 | 3
  Related AE(s) | 4 | 2

17. Secondary Outcome: Number of HIV- Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 4
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 144 | 145
Participants | 1 | 0

18. Secondary Outcome: Number of HIV- Subjects With Medically Significant Conditions (MSCs)
Description: as for outcome 5
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 144 | 145
Participants | 7 | 14

19. Secondary Outcome: Number of HIV- Subjects With Potential Immune-mediated Disease (pIMDs)
Description: as for outcome 6
Time Frame: From Day 0 up to Month 7 (from Day 0 up to 30 days after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 144 | 145
Participants | 0 | 0

20. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: as for outcome 7
Time Frame: During the entire study period (from Day 0 up to Month 24)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 10 | 8 | 3 | 7
Participants
  Live infant NO apparent congenital anomaly | 8 | 7 | 3 | 7
  Live infant congenital anomaly | 0 | 0 | 0 | 0
  Elective termin. NO apparent congenital anomaly | 1 | 0 | 0 | 0
  Elective termin. congenital anomaly | 0 | 0 | 0 | 0
  Ectopic pregnancy | 0 | 0 | 0 | 0
  Spontaneous abortion NO apparent congen. anomaly | 1 | 1 | 0 | 0
  Stillbirth NO apparent congenital anomaly | 0 | 0 | 0 | 0
  Stillbirth congenital anomaly | 0 | 0 | 0 | 0
  Lost to follow-up | 0 | 0 | 0 | 0
  Pregnancy ongoing | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Relevant Abnormalities in Alanine Aminotransferase, Basophils, Creatinine and Eosinophils Parameters
Description: Among assessed haematological and biochemical parameters were: alanine aminotransferase [ALAT], basophils [BSPH], creatinine [CRT], eosinophils [ESPH]. Unknown = value unknown for the specified visit and laboratory parameter; Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 0, Week 6, Week 10, Month 6, Month 7, Month 12, Month 18 and Month 24
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available at Day 0, Week 6, Week 10, Month 6, Month 7*, Month 12, Month 18 and Month 24.
  * Month 7 data for HIV+/Cervarix and HIV+/Gardasil groups are also reported in the Primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants
  ALAT, Day 0, Unknown | 0 | 0 | 0 | 0
  ALAT, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  ALAT, Week 6, Unknown | 0 | 0 | 0 | 0
  ALAT, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  ALAT, Week 10, Unknown | 1 | 0 | 0 | 0
  ALAT, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  ALAT, Month 6, Unknown | 0 | 0 | 0 | 0
  ALAT, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  ALAT, Month 7, Unknown | 0 | 0 | 0 | 0
  ALAT, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  ALAT, Month 12, Unknown | 0 | 0 | 0 | 1
  ALAT, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  ALAT, Month 18, Unknown | 0 | 0 | 0 | 0
  ALAT, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  ALAT, Month 24, Unknown | 0 | 0 | 0 | 0
  ALAT, Day 0, Below | 9 | 4 | 33 | 35
  ALAT, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  ALAT, Week 6, Below | 4 | 5 | 35 | 32
  ALAT, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  ALAT, Week 10, Below | 2 | 8 | 27 | 26
  ALAT, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  ALAT, Month 6, Below | 3 | 4 | 25 | 27
  ALAT, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  ALAT, Month 7, Below | 4 | 3 | 20 | 23
  ALAT, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  ALAT, Month 12, Below | 6 | 1 | 20 | 22
  ALAT, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  ALAT, Month 18, Below | 2 | 2 | 23 | 17
  ALAT, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  ALAT, Month 24, Below | 0 | 1 | 14 | 14
  ALAT, Day 0, Within | 109 | 118 | 109 | 106
  ALAT, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  ALAT, Week 6, Within | 119 | 115 | 97 | 106
  ALAT, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  ALAT, Week 10, Within | 117 | 110 | 104 | 109
  ALAT, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  ALAT, Month 6, Within | 112 | 110 | 101 | 102
  ALAT, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  ALAT, Month 7, Within | 110 | 105 | 94 | 98
  ALAT, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  ALAT, Month 12, Within | 104 | 112 | 86 | 95
  ALAT, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  ALAT, Month 18, Within | 115 | 109 | 85 | 98
  ALAT, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  ALAT, Month 24, Within | 112 | 110 | 87 | 95
  ALAT, Day 0, Above | 11 | 6 | 2 | 4
  ALAT, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  ALAT, Week 6, Above | 5 | 6 | 5 | 4
  ALAT, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  ALAT, Week 10, Above | 8 | 9 | 4 | 1
  ALAT, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  ALAT, Month 6, Above | 8 | 9 | 2 | 5
  ALAT, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  ALAT, Month 7, Above | 7 | 13 | 1 | 4
  ALAT, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  ALAT, Month 12, Above | 12 | 6 | 2 | 0
  ALAT, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  ALAT, Month 18, Above | 4 | 6 | 2 | 2
  ALAT, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  ALAT, Month 24, Above | 4 | 6 | 2 | 2
  BSPH, Day 0, Unknown | 0 | 0 | 0 | 0
  BSPH, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  BSPH, Week 6, Unknown | 0 | 0 | 2 | 3
  BSPH, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  BSPH, Week 10, Unknown | 0 | 0 | 0 | 0
  BSPH, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  BSPH, Month 6, Unknown | 0 | 0 | 0 | 0
  BSPH, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  BSPH, Month 7, Unknown | 0 | 0 | 0 | 0
  BSPH, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  BSPH, Month 12, Unknown | 1 | 0 | 0 | 0
  BSPH, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  BSPH, Month 18, Unknown | 0 | 0 | 0 | 0
  BSPH, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  BSPH, Month 24, Unknown | 1 | 0 | 0 | 0
  BSPH, Day 0, Below | 0 | 1 | 21 | 20
  BSPH, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  BSPH, Week 6, Below | 0 | 1 | 8 | 7
  BSPH, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  BSPH, Week 10, Below | 0 | 0 | 15 | 17
  BSPH, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  BSPH, Month 6, Below | 0 | 0 | 12 | 13
  BSPH, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  BSPH, Month 7, Below | 0 | 0 | 6 | 8
  BSPH, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  BSPH, Month 12, Below | 0 | 0 | 6 | 7
  BSPH, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  BSPH, Month 18, Below | 0 | 0 | 10 | 12
  BSPH, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  BSPH, Month 24, Below | 0 | 0 | 7 | 8
  BSPH, Day 0, Within | 129 | 127 | 123 | 125
  BSPH, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  BSPH, Week 6, Within | 128 | 125 | 127 | 131
  BSPH, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  BSPH, Week 10, Within | 127 | 124 | 119 | 119
  BSPH, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  BSPH, Month 6, Within | 123 | 122 | 116 | 120
  BSPH, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  BSPH, Month 7, Within | 120 | 121 | 109 | 116
  BSPH, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  BSPH, Month 12, Within | 121 | 119 | 102 | 111
  BSPH, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  BSPH, Month 18, Within | 120 | 117 | 99 | 104
  BSPH, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  BSPH, Month 24, Within | 115 | 117 | 96 | 102
  BSPH, Day 0, Above | 0 | 0 | 0 | 0
  BSPH, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  BSPH, Week 6, Above | 0 | 0 | 0 | 1
  BSPH, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  BSPH, Week 10, Above | 1 | 3 | 1 | 0
  BSPH, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  BSPH, Month 6, Above | 0 | 1 | 0 | 1
  BSPH, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  BSPH, Month 7, Above | 1 | 0 | 0 | 1
  BSPH, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  BSPH, Month 12, Above | 0 | 0 | 0 | 0
  BSPH, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  BSPH, Month 18, Above | 1 | 0 | 1 | 1
  BSPH, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  BSPH, Month 24, Above | 0 | 0 | 0 | 1
  CRT, Day 0, Unknown: number analyzed (Participants) | 129 | 127 | 144 | 145
  CRT, Day 0, Unknown | 0 | 0 | 0 | 0
  CRT, Week 6, Unknown: number analyzed (Participants) | 128 | 125 | 137 | 142
  CRT, Week 6, Unknown | 0 | 0 | 0 | 0
  CRT, Week 10, Unknown: number analyzed (Participants) | 128 | 126 | 135 | 136
  CRT, Week 10, Unknown | 0 | 0 | 0 | 0
  CRT, Month 6, Unknown: number analyzed (Participants) | 123 | 122 | 128 | 134
  CRT, Month 6, Unknown | 0 | 0 | 0 | 0
  CRT, Month 7, Unknown: number analyzed (Participants) | 121 | 120 | 115 | 125
  CRT, Month 7, Unknown | 0 | 0 | 0 | 0
  CRT, Month 12, Unknown: number analyzed (Participants) | 122 | 118 | 108 | 118
  CRT, Month 12, Unknown | 0 | 0 | 0 | 0
  CRT, Month 18, Unknown: number analyzed (Participants) | 121 | 116 | 110 | 117
  CRT, Month 18, Unknown | 0 | 0 | 0 | 0
  CRT, Month 24, Unknown: number analyzed (Participants) | 116 | 116 | 103 | 111
  CRT, Month 24, Unknown | 0 | 0 | 0 | 0
  CRT, Day 0, Below: number analyzed (Participants) | 129 | 127 | 144 | 145
  CRT, Day 0, Below | 31 | 26 | 27 | 21
  CRT, Week 6, Below: number analyzed (Participants) | 128 | 125 | 137 | 142
  CRT, Week 6, Below | 35 | 28 | 36 | 28
  CRT, Week 10, Below: number analyzed (Participants) | 128 | 126 | 135 | 136
  CRT, Week 10, Below | 33 | 30 | 27 | 29
  CRT, Month 6, Below: number analyzed (Participants) | 123 | 122 | 128 | 134
  CRT, Month 6, Below | 33 | 32 | 25 | 26
  CRT, Month 7, Below: number analyzed (Participants) | 121 | 120 | 115 | 125
  CRT, Month 7, Below | 29 | 36 | 22 | 17
  CRT, Month 12, Below: number analyzed (Participants) | 122 | 118 | 108 | 118
  CRT, Month 12, Below | 25 | 23 | 24 | 22
  CRT, Month 18, Below: number analyzed (Participants) | 121 | 116 | 110 | 117
  CRT, Month 18, Below | 25 | 17 | 11 | 12
  CRT, Month 24, Below: number analyzed (Participants) | 116 | 116 | 103 | 111
  CRT, Month 24, Below | 27 | 30 | 17 | 17
  CRT, Day 0, Within: number analyzed (Participants) | 129 | 127 | 144 | 145
  CRT, Day 0, Within | 97 | 100 | 115 | 123
  CRT, Week 6, Within: number analyzed (Participants) | 128 | 125 | 137 | 142
  CRT, Week 6, Within | 93 | 97 | 101 | 113
  CRT, Week 10, Within: number analyzed (Participants) | 128 | 126 | 135 | 136
  CRT, Week 10, Within | 95 | 96 | 108 | 107
  CRT, Month 6, Within: number analyzed (Participants) | 123 | 122 | 128 | 134
  CRT, Month 6, Within | 89 | 89 | 103 | 107
  CRT, Month 7, Within: number analyzed (Participants) | 121 | 120 | 115 | 125
  CRT, Month 7, Within | 91 | 84 | 93 | 107
  CRT, Month 12, Within: number analyzed (Participants) | 122 | 118 | 108 | 118
  CRT, Month 12, Within | 94 | 91 | 83 | 95
  CRT, Month 18, Within: number analyzed (Participants) | 121 | 116 | 110 | 117
  CRT, Month 18, Within | 93 | 98 | 98 | 102
  CRT, Month 24, Within: number analyzed (Participants) | 116 | 116 | 103 | 111
  CRT, Month 24, Within | 88 | 85 | 86 | 93
  CRT, Day 0, Above: number analyzed (Participants) | 129 | 127 | 144 | 145
  CRT, Day 0, Above | 1 | 1 | 2 | 1
  CRT, Week 6, Above: number analyzed (Participants) | 128 | 125 | 137 | 142
  CRT, Week 6, Above | 0 | 0 | 0 | 1
  CRT, Week 10, Above: number analyzed (Participants) | 128 | 126 | 135 | 136
  CRT, Week 10, Above | 0 | 0 | 0 | 0
  CRT, Month 6, Above: number analyzed (Participants) | 123 | 122 | 128 | 134
  CRT, Month 6, Above | 1 | 1 | 0 | 1
  CRT, Month 7, Above: number analyzed (Participants) | 121 | 120 | 115 | 125
  CRT, Month 7, Above | 1 | 0 | 0 | 1
  CRT, Month 12, Above: number analyzed (Participants) | 122 | 118 | 108 | 118
  CRT, Month 12, Above | 3 | 4 | 1 | 1
  CRT, Month 18, Above: number analyzed (Participants) | 121 | 116 | 110 | 117
  CRT, Month 18, Above | 3 | 1 | 1 | 3
  CRT, Month 24, Above: number analyzed (Participants) | 116 | 116 | 103 | 111
  CRT, Month 24, Above | 1 | 1 | 0 | 1
  ESPH, Day 0, Unknown | 0 | 0 | 0 | 0
  ESPH, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  ESPH, Week 6, Unknown | 0 | 0 | 2 | 3
  ESPH, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  ESPH, Week 10, Unknown | 0 | 0 | 0 | 0
  ESPH, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  ESPH, Month 6, Unknown | 0 | 0 | 0 | 0
  ESPH, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  ESPH, Month 7, Unknown | 0 | 0 | 0 | 0
  ESPH, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  ESPH, Month 12, Unknown | 1 | 0 | 0 | 0
  ESPH, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  ESPH, Month 18, Unknown | 0 | 0 | 0 | 0
  ESPH, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  ESPH, Month 24, Unknown | 1 | 0 | 0 | 0
  ESPH, Day 0, Below | 15 | 18 | 3 | 4
  ESPH, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  ESPH, Week 6, Below | 10 | 13 | 7 | 6
  ESPH, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  ESPH, Week 10, Below | 11 | 12 | 3 | 1
  ESPH, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  ESPH, Month 6, Below | 9 | 13 | 4 | 4
  ESPH, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  ESPH, Month 7, Below | 9 | 10 | 6 | 6
  ESPH, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  ESPH, Month 12, Below | 9 | 10 | 3 | 6
  ESPH, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  ESPH, Month 18, Below | 4 | 9 | 6 | 4
  ESPH, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  ESPH, Month 24, Below | 7 | 15 | 3 | 6
  ESPH, Day 0, Within | 108 | 102 | 130 | 133
  ESPH, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  ESPH, Week 6, Within | 109 | 102 | 115 | 126
  ESPH, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  ESPH, Week 10, Within | 112 | 108 | 125 | 130
  ESPH, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  ESPH, Month 6, Within | 103 | 108 | 118 | 124
  ESPH, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  ESPH, Month 7, Within | 108 | 106 | 103 | 112
  ESPH, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  ESPH, Month 12, Within | 105 | 104 | 98 | 107
  ESPH, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  ESPH, Month 18, Within | 111 | 106 | 96 | 105
  ESPH, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  ESPH, Month 24, Within | 103 | 99 | 99 | 99
  ESPH, Day 0, Above | 6 | 8 | 11 | 8
  ESPH, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  ESPH, Week 6, Above | 9 | 11 | 13 | 7
  ESPH, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  ESPH, Week 10, Above | 5 | 7 | 7 | 5
  ESPH, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  ESPH, Month 6, Above | 11 | 2 | 6 | 6
  ESPH, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  ESPH, Month 7, Above | 4 | 5 | 6 | 7
  ESPH, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  ESPH, Month 12, Above | 7 | 5 | 7 | 5
  ESPH, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  ESPH, Month 18, Above | 6 | 2 | 8 | 8
  ESPH, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  ESPH, Month 24, Above | 5 | 3 | 1 | 6

22. Secondary Outcome: Number of Subjects With Relevant Abnormalities in Haematocrit, Haemoglobin, Lymphocytes and Monocytes Parameters
Description: Among assessed haematological parameters were: haematocrit [HTCR], haemoglobin [HGB], lymphocytes [LYMP] and monocytes [MONO]. Unknown = value unknown for the specified visit and laboratory parameter; Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 0, Week 6, Week 10, Month 6, Month 7, Month 12, Month 18 and Month 24
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants
  HTCR, Day 0, Unknown | 0 | 0 | 0 | 0
  HTCR, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  HTCR, Week 6, Unknown | 0 | 1 | 0 | 0
  HTCR, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  HTCR, Week 10, Unknown | 0 | 0 | 0 | 0
  HTCR, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  HTCR, Month 6, Unknown | 0 | 0 | 0 | 0
  HTCR, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  HTCR, Month 7, Unknown | 0 | 0 | 0 | 1
  HTCR, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  HTCR, Month 12, Unknown | 1 | 0 | 0 | 0
  HTCR, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  HTCR, Month 18, Unknown | 0 | 0 | 0 | 0
  HTCR, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  HTCR, Month 24, Unknown | 1 | 0 | 0 | 0
  HTCR, Day 0, Below | 32 | 23 | 24 | 24
  HTCR, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  HTCR, Week 6, Below | 22 | 17 | 18 | 13
  HTCR, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  HTCR, Week 10, Below | 30 | 22 | 11 | 7
  HTCR, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  HTCR, Month 6, Below | 26 | 27 | 13 | 17
  HTCR, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  HTCR, Month 7, Below | 19 | 27 | 13 | 14
  HTCR, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  HTCR, Month 12, Below | 24 | 25 | 15 | 17
  HTCR, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  HTCR, Month 18, Below | 30 | 22 | 17 | 16
  HTCR, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  HTCR, Month 24, Below | 24 | 24 | 21 | 17
  HTCR, Day 0, Within | 96 | 102 | 120 | 118
  HTCR, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  HTCR, Week 6, Within | 106 | 105 | 119 | 125
  HTCR, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  HTCR, Week 10, Within | 97 | 103 | 123 | 126
  HTCR, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  HTCR, Month 6, Within | 97 | 95 | 115 | 117
  HTCR, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  HTCR, Month 7, Within | 101 | 92 | 102 | 108
  HTCR, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  HTCR, Month 12, Within | 95 | 94 | 93 | 100
  HTCR, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  HTCR, Month 18, Within | 91 | 92 | 90 | 101
  HTCR, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  HTCR, Month 24, Within | 91 | 92 | 82 | 93
  HTCR, Day 0, Above | 1 | 3 | 0 | 3
  HTCR, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  HTCR, Week 6, Above | 0 | 3 | 0 | 4
  HTCR, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  HTCR, Week 10, Above | 1 | 2 | 1 | 3
  HTCR, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  HTCR, Month 6, Above | 0 | 1 | 0 | 0
  HTCR, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  HTCR, Month 7, Above | 1 | 2 | 0 | 2
  HTCR, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  HTCR, Month 12, Above | 2 | 0 | 0 | 1
  HTCR, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  HTCR, Month 18, Above | 0 | 3 | 3 | 0
  HTCR, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  HTCR, Month 24, Above | 0 | 1 | 0 | 1
  HGB, Day 0, Unknown | 0 | 0 | 0 | 0
  HGB, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  HGB, Week 6, Unknown | 0 | 0 | 0 | 0
  HGB, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  HGB, Week 10, Unknown | 0 | 0 | 0 | 0
  HGB, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  HGB, Month 6, Unknown | 0 | 0 | 0 | 0
  HGB, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  HGB, Month 7, Unknown | 0 | 0 | 0 | 0
  HGB, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  HGB, Month 12, Unknown | 1 | 0 | 0 | 0
  HGB, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  HGB, Month 18, Unknown | 0 | 0 | 0 | 0
  HGB, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  HGB, Month 24, Unknown | 1 | 0 | 0 | 0
  HGB, Day 0, Below | 38 | 37 | 40 | 45
  HGB, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  HGB, Week 6, Below | 38 | 35 | 40 | 50
  HGB, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  HGB, Week 10, Below | 38 | 35 | 37 | 38
  HGB, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  HGB, Month 6, Below | 38 | 36 | 45 | 38
  HGB, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  HGB, Month 7, Below | 28 | 37 | 36 | 38
  HGB, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  HGB, Month 12, Below | 29 | 35 | 39 | 39
  HGB, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  HGB, Month 18, Below | 34 | 32 | 32 | 35
  HGB, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  HGB, Month 24, Below | 27 | 27 | 28 | 26
  HGB, Day 0, Within | 88 | 89 | 104 | 98
  HGB, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  HGB, Week 6, Within | 88 | 88 | 97 | 88
  HGB, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  HGB, Week 10, Within | 89 | 90 | 98 | 97
  HGB, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  HGB, Month 6, Within | 85 | 86 | 83 | 96
  HGB, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  HGB, Month 7, Within | 92 | 83 | 79 | 86
  HGB, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  HGB, Month 12, Within | 91 | 83 | 69 | 79
  HGB, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  HGB, Month 18, Within | 84 | 82 | 77 | 82
  HGB, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  HGB, Month 24, Within | 88 | 89 | 75 | 84
  HGB, Day 0, Above | 3 | 2 | 0 | 2
  HGB, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  HGB, Week 6, Above | 2 | 3 | 0 | 4
  HGB, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  HGB, Week 10, Above | 1 | 2 | 0 | 1
  HGB, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  HGB, Month 6, Above | 0 | 1 | 0 | 0
  HGB, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  HGB, Month 7, Above | 1 | 1 | 0 | 1
  HGB, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  HGB, Month 12, Above | 1 | 1 | 0 | 0
  HGB, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  HGB, Month 18, Above | 3 | 3 | 1 | 0
  HGB, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  HGB, Month 24, Above | 0 | 1 | 0 | 1
  LYMP, Day 0, Unknown | 0 | 0 | 0 | 0
  LYMP, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  LYMP, Week 6, Unknown | 0 | 0 | 2 | 3
  LYMP, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  LYMP, Week 10, Unknown | 0 | 0 | 0 | 0
  LYMP, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  LYMP, Month 6, Unknown | 0 | 0 | 0 | 0
  LYMP, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  LYMP, Month 7, Unknown | 0 | 0 | 0 | 0
  LYMP, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  LYMP, Month 12, Unknown | 1 | 0 | 0 | 0
  LYMP, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  LYMP, Month 18, Unknown | 0 | 0 | 0 | 0
  LYMP, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  LYMP, Month 24, Unknown | 1 | 0 | 0 | 0
  LYMP, Day 0, Below | 7 | 9 | 11 | 6
  LYMP, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  LYMP, Week 6, Below | 6 | 11 | 12 | 6
  LYMP, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  LYMP, Week 10, Below | 11 | 9 | 13 | 6
  LYMP, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  LYMP, Month 6, Below | 6 | 8 | 9 | 11
  LYMP, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  LYMP, Month 7, Below | 12 | 11 | 6 | 6
  LYMP, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  LYMP, Month 12, Below | 6 | 10 | 6 | 8
  LYMP, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  LYMP, Month 18, Below | 4 | 4 | 6 | 4
  LYMP, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  LYMP, Month 24, Below | 8 | 9 | 6 | 7
  LYMP, Day 0, Within | 105 | 105 | 120 | 132
  LYMP, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  LYMP, Week 6, Within | 109 | 109 | 113 | 121
  LYMP, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  LYMP, Week 10, Within | 101 | 102 | 110 | 124
  LYMP, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  LYMP, Month 6, Within | 98 | 104 | 106 | 115
  LYMP, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  LYMP, Month 7, Within | 96 | 97 | 103 | 111
  LYMP, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  LYMP, Month 12, Within | 104 | 95 | 92 | 98
  LYMP, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  LYMP, Month 18, Within | 105 | 103 | 94 | 106
  LYMP, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  LYMP, Month 24, Within | 98 | 97 | 88 | 101
  LYMP, Day 0, Above | 17 | 14 | 13 | 7
  LYMP, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  LYMP, Week 6, Above | 13 | 6 | 10 | 12
  LYMP, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  LYMP, Week 10, Above | 16 | 16 | 12 | 6
  LYMP, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  LYMP, Month 6, Above | 19 | 11 | 13 | 8
  LYMP, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  LYMP, Month 7, Above | 13 | 13 | 6 | 8
  LYMP, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  LYMP, Month 12, Above | 11 | 14 | 10 | 12
  LYMP, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  LYMP, Month 18, Above | 12 | 10 | 10 | 7
  LYMP, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  LYMP, Month 24, Above | 9 | 11 | 9 | 3
  MONO, Day 0, Unknown | 0 | 0 | 0 | 0
  MONO, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  MONO, Week 6, Unknown | 0 | 0 | 2 | 3
  MONO, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  MONO, Week 10, Unknown | 0 | 0 | 0 | 0
  MONO, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  MONO, Month 6, Unknown | 0 | 0 | 0 | 0
  MONO, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  MONO, Month 7, Unknown | 0 | 0 | 0 | 0
  MONO, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  MONO, Month 12, Unknown | 1 | 0 | 0 | 0
  MONO, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  MONO, Month 18, Unknown | 0 | 0 | 0 | 0
  MONO, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  MONO, Month 24, Unknown | 1 | 0 | 0 | 0
  MONO, Day 0, Below | 7 | 4 | 10 | 17
  MONO, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  MONO, Week 6, Below | 4 | 4 | 3 | 4
  MONO, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  MONO, Week 10, Below | 4 | 4 | 2 | 6
  MONO, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  MONO, Month 6, Below | 3 | 5 | 0 | 7
  MONO, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  MONO, Month 7, Below | 4 | 7 | 5 | 2
  MONO, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  MONO, Month 12, Below | 2 | 5 | 5 | 2
  MONO, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  MONO, Month 18, Below | 3 | 6 | 5 | 4
  MONO, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  MONO, Month 24, Below | 5 | 5 | 7 | 10
  MONO, Day 0, Within | 111 | 117 | 133 | 126
  MONO, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  MONO, Week 6, Within | 117 | 112 | 129 | 133
  MONO, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  MONO, Week 10, Within | 116 | 108 | 129 | 127
  MONO, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  MONO, Month 6, Within | 107 | 104 | 113 | 121
  MONO, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  MONO, Month 7, Within | 106 | 97 | 107 | 118
  MONO, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  MONO, Month 12, Within | 104 | 101 | 101 | 113
  MONO, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  MONO, Month 18, Within | 108 | 99 | 101 | 109
  MONO, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  MONO, Month 24, Within | 98 | 99 | 95 | 99
  MONO, Day 0, Above | 11 | 7 | 1 | 2
  MONO, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  MONO, Week 6, Above | 7 | 10 | 3 | 2
  MONO, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  MONO, Week 10, Above | 8 | 15 | 4 | 3
  MONO, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  MONO, Month 6, Above | 13 | 14 | 6 | 6
  MONO, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  MONO, Month 7, Above | 11 | 17 | 3 | 5
  MONO, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  MONO, Month 12, Above | 15 | 13 | 2 | 3
  MONO, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  MONO, Month 18, Above | 10 | 12 | 4 | 4
  MONO, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  MONO, Month 24, Above | 12 | 13 | 1 | 2

23. Secondary Outcome: Number of Subjects With Relevant Abnormalities in Neutrophils, Platelets, Red Blood Cells and White Blood Cells Parameters
Description: Among assessed haematological parameters were: neutrophils [NTPH], platelets [PLAT], red blood cells [RBC] and white blood cells [WBC]. Unknown = value unknown for the specified visit and laboratory parameter; Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 0, Week 6, Week 10, Month 6, Month 7, Month 12, Month 18 and Month 24
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants
  NTPH, Day 0, Unknown | 0 | 0 | 0 | 0
  NTPH, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  NTPH, Week 6, Unknown | 0 | 0 | 2 | 3
  NTPH, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  NTPH, Week 10, Unknown | 0 | 0 | 0 | 0
  NTPH, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  NTPH, Month 6, Unknown | 0 | 0 | 0 | 0
  NTPH, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  NTPH, Month 7, Unknown | 0 | 0 | 0 | 0
  NTPH, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  NTPH, Month 12, Unknown | 1 | 0 | 0 | 0
  NTPH, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  NTPH, Month 18, Unknown | 0 | 0 | 0 | 0
  NTPH, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  NTPH, Month 24, Unknown | 1 | 0 | 0 | 0
  NTPH, Day 0, Below | 14 | 12 | 11 | 7
  NTPH, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  NTPH, Week 6, Below | 16 | 13 | 8 | 13
  NTPH, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  NTPH, Week 10, Below | 18 | 17 | 12 | 10
  NTPH, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  NTPH, Month 6, Below | 18 | 14 | 15 | 14
  NTPH, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  NTPH, Month 7, Below | 16 | 17 | 10 | 9
  NTPH, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  NTPH, Month 12, Below | 19 | 16 | 12 | 11
  NTPH, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  NTPH, Month 18, Below | 15 | 15 | 9 | 14
  NTPH, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  NTPH, Month 24, Below | 14 | 11 | 9 | 10
  NTPH, Day 0, Within | 106 | 99 | 117 | 122
  NTPH, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  NTPH, Week 6, Within | 101 | 95 | 107 | 116
  NTPH, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  NTPH, Week 10, Within | 103 | 100 | 104 | 113
  NTPH, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  NTPH, Month 6, Within | 100 | 98 | 98 | 104
  NTPH, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  NTPH, Month 7, Within | 97 | 93 | 92 | 106
  NTPH, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  NTPH, Month 12, Within | 92 | 93 | 84 | 94
  NTPH, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  NTPH, Month 18, Within | 98 | 89 | 86 | 92
  NTPH, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  NTPH, Month 24, Within | 92 | 95 | 83 | 89
  NTPH, Day 0, Above | 9 | 17 | 16 | 16
  NTPH, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  NTPH, Week 6, Above | 11 | 18 | 20 | 10
  NTPH, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  NTPH, Week 10, Above | 7 | 10 | 19 | 13
  NTPH, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  NTPH, Month 6, Above | 5 | 11 | 15 | 16
  NTPH, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  NTPH, Month 7, Above | 8 | 11 | 13 | 10
  NTPH, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  NTPH, Month 12, Above | 10 | 10 | 12 | 13
  NTPH, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  NTPH, Month 18, Above | 8 | 13 | 15 | 11
  NTPH, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  NTPH, Month 24, Above | 9 | 11 | 11 | 12
  PLAT, Day 0, Unknown | 0 | 0 | 0 | 0
  PLAT, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 137 | 142
  PLAT, Week 6, Unknown | 0 | 0 | 1 | 1
  PLAT, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 135 | 136
  PLAT, Week 10, Unknown | 0 | 0 | 1 | 0
  PLAT, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 128 | 134
  PLAT, Month 6, Unknown | 0 | 0 | 0 | 0
  PLAT, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  PLAT, Month 7, Unknown | 0 | 0 | 1 | 0
  PLAT, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  PLAT, Month 12, Unknown | 1 | 0 | 1 | 0
  PLAT, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 117
  PLAT, Month 18, Unknown | 0 | 0 | 0 | 0
  PLAT, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  PLAT, Month 24, Unknown | 1 | 0 | 0 | 0
  PLAT, Day 0, Below | 0 | 0 | 3 | 0
  PLAT, Week 6, Below: number analyzed (Participants) | 128 | 126 | 137 | 142
  PLAT, Week 6, Below | 1 | 0 | 1 | 0
  PLAT, Week 10, Below: number analyzed (Participants) | 128 | 127 | 135 | 136
  PLAT, Week 10, Below | 1 | 1 | 0 | 0
  PLAT, Month 6, Below: number analyzed (Participants) | 123 | 123 | 128 | 134
  PLAT, Month 6, Below | 2 | 2 | 0 | 0
  PLAT, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  PLAT, Month 7, Below | 1 | 3 | 1 | 1
  PLAT, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  PLAT, Month 12, Below | 3 | 1 | 0 | 2
  PLAT, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 117
  PLAT, Month 18, Below | 3 | 4 | 1 | 2
  PLAT, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  PLAT, Month 24, Below | 1 | 2 | 2 | 3
  PLAT, Day 0, Within | 123 | 122 | 133 | 138
  PLAT, Week 6, Within: number analyzed (Participants) | 128 | 126 | 137 | 142
  PLAT, Week 6, Within | 124 | 119 | 130 | 137
  PLAT, Week 10, Within: number analyzed (Participants) | 128 | 127 | 135 | 136
  PLAT, Week 10, Within | 122 | 124 | 131 | 132
  PLAT, Month 6, Within: number analyzed (Participants) | 123 | 123 | 128 | 134
  PLAT, Month 6, Within | 116 | 118 | 127 | 131
  PLAT, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  PLAT, Month 7, Within | 118 | 114 | 110 | 121
  PLAT, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  PLAT, Month 12, Within | 113 | 114 | 103 | 111
  PLAT, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 117
  PLAT, Month 18, Within | 117 | 110 | 106 | 111
  PLAT, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  PLAT, Month 24, Within | 109 | 110 | 97 | 103
  PLAT, Day 0, Above | 6 | 6 | 8 | 7
  PLAT, Week 6, Above: number analyzed (Participants) | 128 | 126 | 137 | 142
  PLAT, Week 6, Above | 3 | 7 | 5 | 4
  PLAT, Week 10, Above: number analyzed (Participants) | 128 | 127 | 135 | 136
  PLAT, Week 10, Above | 5 | 2 | 3 | 4
  PLAT, Month 6, Above: number analyzed (Participants) | 123 | 123 | 128 | 134
  PLAT, Month 6, Above | 5 | 3 | 1 | 3
  PLAT, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  PLAT, Month 7, Above | 2 | 4 | 3 | 3
  PLAT, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  PLAT, Month 12, Above | 5 | 4 | 4 | 5
  PLAT, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 117
  PLAT, Month 18, Above | 1 | 3 | 3 | 4
  PLAT, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  PLAT, Month 24, Above | 5 | 5 | 4 | 5
  RBC, Day 0, Unknown: number analyzed (Participants) | 129 | 128 | 141 | 141
  RBC, Day 0, Unknown | 0 | 0 | 0 | 0
  RBC, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 136 | 139
  RBC, Week 6, Unknown | 0 | 0 | 0 | 1
  RBC, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 134 | 135
  RBC, Week 10, Unknown | 0 | 0 | 0 | 0
  RBC, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 127 | 134
  RBC, Month 6, Unknown | 0 | 0 | 0 | 1
  RBC, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 115 | 125
  RBC, Month 7, Unknown | 0 | 0 | 0 | 0
  RBC, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 108 | 118
  RBC, Month 12, Unknown | 1 | 0 | 0 | 1
  RBC, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 110 | 116
  RBC, Month 18, Unknown | 0 | 0 | 2 | 3
  RBC, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 103 | 111
  RBC, Month 24, Unknown | 1 | 0 | 0 | 0
  RBC, Day 0, Below: number analyzed (Participants) | 129 | 128 | 141 | 141
  RBC, Day 0, Below | 43 | 38 | 18 | 13
  RBC, Week 6, Below: number analyzed (Participants) | 128 | 126 | 136 | 139
  RBC, Week 6, Below | 44 | 36 | 14 | 12
  RBC, Week 10, Below: number analyzed (Participants) | 128 | 127 | 134 | 135
  RBC, Week 10, Below | 48 | 37 | 11 | 8
  RBC, Month 6, Below: number analyzed (Participants) | 123 | 123 | 127 | 134
  RBC, Month 6, Below | 40 | 39 | 14 | 12
  RBC, Month 7, Below: number analyzed (Participants) | 121 | 121 | 115 | 125
  RBC, Month 7, Below | 36 | 34 | 15 | 19
  RBC, Month 12, Below: number analyzed (Participants) | 122 | 119 | 108 | 118
  RBC, Month 12, Below | 39 | 31 | 19 | 14
  RBC, Month 18, Below: number analyzed (Participants) | 121 | 117 | 110 | 116
  RBC, Month 18, Below | 38 | 31 | 9 | 13
  RBC, Month 24, Below: number analyzed (Participants) | 116 | 117 | 103 | 111
  RBC, Month 24, Below | 38 | 34 | 10 | 9
  RBC, Day 0, Within: number analyzed (Participants) | 129 | 128 | 141 | 141
  RBC, Day 0, Within | 83 | 87 | 118 | 123
  RBC, Week 6, Within: number analyzed (Participants) | 128 | 126 | 136 | 139
  RBC, Week 6, Within | 81 | 85 | 118 | 120
  RBC, Week 10, Within: number analyzed (Participants) | 128 | 127 | 134 | 135
  RBC, Week 10, Within | 78 | 87 | 120 | 122
  RBC, Month 6, Within: number analyzed (Participants) | 123 | 123 | 127 | 134
  RBC, Month 6, Within | 79 | 81 | 111 | 117
  RBC, Month 7, Within: number analyzed (Participants) | 121 | 121 | 115 | 125
  RBC, Month 7, Within | 82 | 84 | 100 | 100
  RBC, Month 12, Within: number analyzed (Participants) | 122 | 119 | 108 | 118
  RBC, Month 12, Within | 79 | 86 | 88 | 100
  RBC, Month 18, Within: number analyzed (Participants) | 121 | 117 | 110 | 116
  RBC, Month 18, Within | 81 | 80 | 97 | 96
  RBC, Month 24, Within: number analyzed (Participants) | 116 | 117 | 103 | 111
  RBC, Month 24, Within | 74 | 83 | 91 | 98
  RBC, Day 0, Above: number analyzed (Participants) | 129 | 128 | 141 | 141
  RBC, Day 0, Above | 3 | 3 | 5 | 5
  RBC, Week 6, Above: number analyzed (Participants) | 128 | 126 | 136 | 139
  RBC, Week 6, Above | 3 | 5 | 4 | 6
  RBC, Week 10, Above: number analyzed (Participants) | 128 | 127 | 134 | 135
  RBC, Week 10, Above | 2 | 3 | 3 | 5
  RBC, Month 6, Above: number analyzed (Participants) | 123 | 123 | 127 | 134
  RBC, Month 6, Above | 4 | 3 | 2 | 4
  RBC, Month 7, Above: number analyzed (Participants) | 121 | 121 | 115 | 125
  RBC, Month 7, Above | 3 | 3 | 0 | 6
  RBC, Month 12, Above: number analyzed (Participants) | 122 | 119 | 108 | 118
  RBC, Month 12, Above | 3 | 2 | 1 | 3
  RBC, Month 18, Above: number analyzed (Participants) | 121 | 117 | 110 | 116
  RBC, Month 18, Above | 2 | 6 | 2 | 4
  RBC, Month 24, Above: number analyzed (Participants) | 116 | 117 | 103 | 111
  RBC, Month 24, Above | 3 | 0 | 2 | 4
  WBC, Day 0, Unknown: number analyzed (Participants) | 129 | 128 | 143 | 145
  WBC, Day 0, Unknown | 0 | 0 | 0 | 0
  WBC, Week 6, Unknown: number analyzed (Participants) | 128 | 126 | 136 | 142
  WBC, Week 6, Unknown | 0 | 0 | 0 | 0
  WBC, Week 10, Unknown: number analyzed (Participants) | 128 | 127 | 134 | 136
  WBC, Week 10, Unknown | 0 | 0 | 0 | 0
  WBC, Month 6, Unknown: number analyzed (Participants) | 123 | 123 | 127 | 134
  WBC, Month 6, Unknown | 0 | 0 | 0 | 0
  WBC, Month 7, Unknown: number analyzed (Participants) | 121 | 121 | 114 | 125
  WBC, Month 7, Unknown | 0 | 0 | 0 | 0
  WBC, Month 12, Unknown: number analyzed (Participants) | 122 | 119 | 107 | 118
  WBC, Month 12, Unknown | 1 | 0 | 0 | 0
  WBC, Month 18, Unknown: number analyzed (Participants) | 121 | 117 | 109 | 117
  WBC, Month 18, Unknown | 0 | 0 | 0 | 0
  WBC, Month 24, Unknown: number analyzed (Participants) | 116 | 117 | 102 | 111
  WBC, Month 24, Unknown | 1 | 0 | 0 | 0
  WBC, Day 0, Below: number analyzed (Participants) | 129 | 128 | 143 | 145
  WBC, Day 0, Below | 8 | 7 | 5 | 2
  WBC, Week 6, Below: number analyzed (Participants) | 128 | 126 | 136 | 142
  WBC, Week 6, Below | 9 | 11 | 5 | 4
  WBC, Week 10, Below: number analyzed (Participants) | 128 | 127 | 134 | 136
  WBC, Week 10, Below | 9 | 9 | 2 | 3
  WBC, Month 6, Below: number analyzed (Participants) | 123 | 123 | 127 | 134
  WBC, Month 6, Below | 12 | 6 | 2 | 2
  WBC, Month 7, Below: number analyzed (Participants) | 121 | 121 | 114 | 125
  WBC, Month 7, Below | 10 | 9 | 5 | 1
  WBC, Month 12, Below: number analyzed (Participants) | 122 | 119 | 107 | 118
  WBC, Month 12, Below | 14 | 13 | 3 | 2
  WBC, Month 18, Below: number analyzed (Participants) | 121 | 117 | 109 | 117
  WBC, Month 18, Below | 12 | 10 | 4 | 5
  WBC, Month 24, Below: number analyzed (Participants) | 116 | 117 | 102 | 111
  WBC, Month 24, Below | 11 | 5 | 3 | 4
  WBC, Day 0, Within: number analyzed (Participants) | 129 | 128 | 143 | 145
  WBC, Day 0, Within | 118 | 116 | 135 | 140
  WBC, Week 6, Within: number analyzed (Participants) | 128 | 126 | 136 | 142
  WBC, Week 6, Within | 118 | 111 | 124 | 135
  WBC, Week 10, Within: number analyzed (Participants) | 128 | 127 | 134 | 136
  WBC, Week 10, Within | 116 | 113 | 131 | 129
  WBC, Month 6, Within: number analyzed (Participants) | 123 | 123 | 127 | 134
  WBC, Month 6, Within | 106 | 116 | 122 | 128
  WBC, Month 7, Within: number analyzed (Participants) | 121 | 121 | 114 | 125
  WBC, Month 7, Within | 106 | 108 | 106 | 120
  WBC, Month 12, Within: number analyzed (Participants) | 122 | 119 | 107 | 118
  WBC, Month 12, Within | 103 | 103 | 100 | 115
  WBC, Month 18, Within: number analyzed (Participants) | 121 | 117 | 109 | 117
  WBC, Month 18, Within | 106 | 107 | 100 | 107
  WBC, Month 24, Within: number analyzed (Participants) | 116 | 117 | 102 | 111
  WBC, Month 24, Within | 102 | 107 | 94 | 101
  WBC, Day 0, Above: number analyzed (Participants) | 129 | 128 | 143 | 145
  WBC, Day 0, Above | 3 | 5 | 3 | 3
  WBC, Week 6, Above: number analyzed (Participants) | 128 | 126 | 136 | 142
  WBC, Week 6, Above | 1 | 4 | 7 | 3
  WBC, Week 10, Above: number analyzed (Participants) | 128 | 127 | 134 | 136
  WBC, Week 10, Above | 3 | 5 | 1 | 4
  WBC, Month 6, Above: number analyzed (Participants) | 123 | 123 | 127 | 134
  WBC, Month 6, Above | 5 | 1 | 3 | 4
  WBC, Month 7, Above: number analyzed (Participants) | 121 | 121 | 114 | 125
  WBC, Month 7, Above | 5 | 4 | 3 | 4
  WBC, Month 12, Above: number analyzed (Participants) | 122 | 119 | 107 | 118
  WBC, Month 12, Above | 4 | 3 | 4 | 1
  WBC, Month 18, Above: number analyzed (Participants) | 121 | 117 | 109 | 117
  WBC, Month 18, Above | 3 | 0 | 5 | 5
  WBC, Month 24, Above: number analyzed (Participants) | 116 | 117 | 102 | 111
  WBC, Month 24, Above | 2 | 5 | 5 | 6

24. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 4
Time Frame: During the entire study period (from Day 0 up to Month 24)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants | 9 | 9 | 4 | 1

25. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs)
Description: as for outcome 5
Time Frame: From Day 0 up to Month 18 (from Day 0 up to 12 months after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants | 25 | 37 | 10 | 17

26. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 6
Time Frame: From Day 0 up to Month 18 (from Day 0 up to 12 months after the last vaccination dose at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 129 | 128 | 144 | 145
Participants | 1 | 0 | 0 | 0

27. Secondary Outcome: Cluster of Differentiation 4 (CD4+) Cell Count in HIV+ Subjects at Months 12, 18 and 24
Description: CD4+ cell count, expressed in cells/cubic millimeter (mm3), was assessed for HIV+ subjects.
Time Frame: At Months 12, 18 and 24
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available at Months 12, 18 and 24.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 122 | 119
cells/mm3
  CD4+ cell counts, Month 12 | 584.5 [498.0 to 832.0] | 602.0 [445.0 to 835.0]
  CD4+ cell counts, Month 18: number analyzed (Participants) | 121 | 117
  CD4+ cell counts, Month 18 | 621.0 [472.0 to 789.0] | 572.0 [443.0 to 770.0]
  CD4+ cell counts, Month 24: number analyzed (Participants) | 115 | 117
  CD4+ cell counts, Month 24 | 568.0 [447.0 to 738.0] | 598.0 [441.0 to 834.0]

28. Secondary Outcome: HIV Viral Load (VL) in HIV+ Subjects at Months 12, 18 and 24
Description: HIV VL, expressed in HIV copies/milliliter (mL), was assessed for HIV+ subjects.
Time Frame: At Months 12, 18 and 24
Population: as for outcome 27
Measure: Median (Inter-Quartile Range); unit: HIV copies/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 94 | 96
HIV copies/mL
  HIV viral load, Month 12 | 1.6 [1.3 to 3.2] | 2.3 [1.3 to 3.7]
  HIV viral load, Month 18: number analyzed (Participants) | 94 | 91
  HIV viral load, Month 18 | 1.7 [1.3 to 3.2] | 2.2 [1.3 to 3.8]
  HIV viral load, Month 24: number analyzed (Participants) | 93 | 87
  HIV viral load, Month 24 | 1.6 [1.3 to 2.8] | 2.1 [1.3 to 3.8]

29. Secondary Outcome: Number of HIV+ Subjects by WHO HIV Clinical Staging
Description: HIV+ subjects were categorised into clinical stages 1 through 4, as per the WHO classification [WHO, 2009].
Time Frame: At Months 12, 18 and 24
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group
Number analyzed (Participants) | 129 | 128
Participants
  Clinical stage 1, Month 12 | 113 | 112
  Clinical stage 2, Month 12 | 7 | 1
  Clinical stage 3, Month 12 | 1 | 2
  Clinical stage 4, Month 12 | 2 | 4
  Clinical stage 1, Month 18 | 112 | 110
  Clinical stage 2, Month 18 | 7 | 1
  Clinical stage 3, Month 18 | 1 | 2
  Clinical stage 4, Month 18 | 2 | 4
  Clinical stage 1, Month 24 | 107 | 110
  Clinical stage 2, Month 24 | 7 | 1
  Clinical stage 3, Month 24 | 1 | 2
  Clinical stage 4, Month 24 | 2 | 4

30. Secondary Outcome: Pseudovirion-Based Neutralization Assay (PBNA) Titers of Anti-HPV-16/18 Antibodies in HIV- Subjects, Based on TVC
Description: Titers of anti-HPV-16/18 antibodies, expressed as Geometric Mean Titers (GMTs), with cut-offs greater than or equal to (≥) 40 estimated dose giving 50% signal reduction when compared to a control without serum (ED50), as assessed by the Pseudovirion-Based Neutralization Assay [PBNA], for HIV- subjects.
  Between-group comparisons to assess superiority were performed on the TVC (by PBNA, regardless of HPV serostatus at baseline).
Time Frame: At Month 7 (30 days after the last vaccination dose at Month 6)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 105 | 112
Titers
  Anti-HPV-16 | 60550.6 [44040.1 to 83250.9] | 19634.8 [14410.8 to 26752.4]
  Anti-HPV-18: number analyzed (Participants) | 105 | 111
  Anti-HPV-18 | 32118.1 [23195.8 to 44472.3] | 5773.4 [4205.2 to 7926.4]
Statistical Analysis 1: Comparison: HIV-/Cervarix Group vs HIV-/Gardasil Group; Adjusted GMT ratio for anti-HPV-18 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV-/Cervarix Group) was superior to that of Gardasil vaccine (HIV-/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-18, measured by Pseudovirion-based neutralization assay (PBNA) in HIV- subjects; Test type: Superiority — Superiority was defined as the lower limit of the 97.5% CI for the ratio of GMTs (Cervarix over Gardasil) for HPV-18 type being above 1, with a statistically significant p-value; p < 0.0001, ANOVA; ANOVA model on the log10 transformation of the titers for HIV- subjects and including the vaccine group as fixed effect; Adjusted GMT ratio = 5.38, 97.5% CI 2-sided [3.20 to 9.06]
Statistical Analysis 2: Comparison: HIV-/Cervarix Group vs HIV-/Gardasil Group; Adjusted GMT ratio for anti-HPV-16 neutra antibody (ED50): To demonstrate that the immunogenicity of Cervarix vaccine (HIV-/Cervarix Group) was superior to that of Gardasil vaccine (HIV-/Gardasil Group), in terms of geometric mean titers (GMTs) against HPV-16, measured by Pseudovirion-based neutralization assay (PBNA) in HIV- subjects; Test type: Superiority — Superiority was defined as the lower limit of the 97.5% CI for the ratio of GMTs (Cervarix over Gardasil) for HPV-16 type being above 1, with a statistically significant p-value; p < 0.0001, ANOVA; ANOVA model on the log10 transformation of the titers for HIV- subjects and including the vaccine group as fixed effect; Adjusted GMT ratio = 3.05, 97.5% CI 2-sided [1.84 to 5.06]

31. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations by Enzyme-linked Immunosorbent Assay (ELISA) in Serum
Description: Anti-HPV-16 and anti-HPV-18 antibody concentrations in serum, are presented as Geometric Mean Concentrations (GMCs), with cut-offs greater than or equal to (≥) 19 ELISA units per milliliter (EU/mL) and 18 EU/mL respectively, as assessed by Enzyme-linked immunosorbent assay (ELISA), in all (HIV+ and HIV-) subjects.
Time Frame: At Day 0, Week 6, Week 10, Month 7, Month 12, Month 18 and Month 24
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity corresponding to each time point were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 81 | 84 | 77 | 80
EU/mL
  anti-HPV-16, Day 0 | 17.2 [13.3 to 22.2] | 15.0 [12.0 to 18.9] | 10.2 [9.4 to 11.0] | 10.9 [9.5 to 12.5]
  anti-HPV-16, Week 6 | 452.9 [302.3 to 678.5] | 280.2 [182.5 to 430.1] | 390.6 [298.3 to 511.6] | 303.2 [228.0 to 403.3]
  anti-HPV-16, Week 10 | 2191.2 [1775.7 to 2704.0] | 1565.5 [1197.5 to 2046.6] | 4512.7 [3771.5 to 5399.7] | 2993.2 [2459.1 to 3643.3]
  anti-HPV-16, Month 7 | 4896.0 [4002.2 to 5989.3] | 2145.2 [1647.8 to 2792.7] | 15493.0 [12537.0 to 19146.0] | 5960.9 [5028.9 to 7065.7]
  anti-HPV-16, Month 12: number analyzed (Participants) | 81 | 81 | 73 | 76
  anti-HPV-16, Month 12 | 1392.3 [1077.5 to 1799.0] | 608.8 [445.4 to 832.1] | 4389.3 [3400.5 to 5665.7] | 1772.2 [1473.3 to 2131.7]
  anti-HPV-16, Month 18: number analyzed (Participants) | 77 | 76 | 70 | 72
  anti-HPV-16, Month 18 | 861.3 [662.3 to 1119.9] | 311.4 [226.3 to 428.4] | 2294.1 [1785.0 to 2948.4] | 798.0 [646.6 to 984.8]
  anti-HPV-16, Month 24: number analyzed (Participants) | 71 | 74 | 64 | 69
  anti-HPV-16, Month 24 | 664.6 [499.9 to 883.7] | 243.5 [173.9 to 341.0] | 1893.6 [1443.8 to 2483.7] | 601.9 [481.8 to 752.1]
  anti-HPV-18, Day 0 | 13.4 [11.2 to 16.0] | 10.7 [9.3 to 12.3] | 9.3 [8.9 to 9.8] | 9.2 [8.9 to 9.5]
  anti-HPV-18, Week 6 | 205.6 [146.3 to 288.7] | 53.2 [36.4 to 77.6] | 277.3 [217.5 to 353.5] | 60.4 [47.5 to 76.8]
  anti-HPV-18, Week 10 | 1432.4 [1136.9 to 1804.6] | 277.2 [200.8 to 382.8] | 3174.4 [2596.2 to 3881.4] | 666.1 [549.8 to 806.9]
  anti-HPV-18, Month 7 | 2540.8 [2085.9 to 3094.9] | 493.8 [356.6 to 683.8] | 6779.3 [5382.6 to 8538.5] | 1516.5 [1232.9 to 1865.2]
  anti-HPV-18, Month 12: number analyzed (Participants) | 81 | 81 | 73 | 76
  anti-HPV-18, Month 12 | 676.9 [520.1 to 880.9] | 116.2 [82.2 to 164.2] | 1747.7 [1329.4 to 2297.6] | 338.3 [261.2 to 438.1]
  anti-HPV-18, Month 18: number analyzed (Participants) | 77 | 76 | 70 | 72
  anti-HPV-18, Month 18 | 408.7 [310.4 to 538.2] | 55.6 [39.6 to 78.0] | 895.5 [679.6 to 1179.9] | 160.1 [123.7 to 207.1]
  anti-HPV-18, Month 24: number analyzed (Participants) | 71 | 74 | 64 | 69
  anti-HPV-18, Month 24 | 295.2 [216.9 to 401.7] | 52.4 [37.2 to 73.8] | 761.9 [576.6 to 1006.7] | 116.2 [88.8 to 151.9]

32. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations by ELISA in Cervicovaginal Secretion (CVS)
Description: Anti-HPV-16 and anti-HPV-18 antibody concentrations in CVS, are presented as Geometric Mean Concentrations (GMCs), with cut-offs greater than or equal to (≥) 0 EU/mL, as assessed by ELISA, in post-menarcheal subjects who volunteered for this procedure.
Time Frame: At Day 0, Week 6, Week 10, Month 7, Month 12, Month 18 and Month 24
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity, which included post-menarcheal subjects who volunteered for this procedure, met all eligibility criteria and for whom data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity corresponding to each time point were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 12 | 18 | 3 | 5
EU/mL
  anti-HPV-16, Day 0 | 1.5 [0.8 to 2.6] | 1.4 [0.7 to 2.8] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  anti-HPV-16, Week 6: number analyzed (Participants) | 7 | 11 | 3 | 5
  anti-HPV-16, Week 6 | 31.5 [4.7 to 211.5] | 3.1 [0.8 to 11.6] | 27.1 [8.7 to 84.2] | 2.7 [0.4 to 16.5]
  anti-HPV-16, Week 10: number analyzed (Participants) | 9 | 11 | 0 | 1
  anti-HPV-16, Week 10 | 38.8 [6.1 to 245.0] | 15.7 [5.4 to 45.2] |  | 159.8 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.
  anti-HPV-16, Month 7: number analyzed (Participants) | 8 | 14 | 3 | 3
  anti-HPV-16, Month 7 | 23.6 [3.4 to 163.0] | 5.4 [1.6 to 17.6] | 104.2 [40.3 to 269.4] | 53.5 [3.0 to 945.1]
  anti-HPV-16, Month 12: number analyzed (Participants) | 9 | 15 | 2 | 1
  anti-HPV-16, Month 12 | 18.7 [3.2 to 109.0] | 6.8 [2.1 to 22.3] | 107.6 [29.1 to 398.1] | 34.7 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.
  anti-HPV-16, Month 24: number analyzed (Participants) | 7 | 10 | 3 | 1
  anti-HPV-16, Month 24 | 8.1 [1.3 to 50.3] | 4.3 [1.4 to 12.9] | 49.0 [4.5 to 534.2] | 1.0 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.
  anti-HPV-18, Day 0 | 1.2 [0.8 to 1.9] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  anti-HPV-18, Week 6: number analyzed (Participants) | 7 | 11 | 3 | 5
  anti-HPV-18, Week 6 | 16.8 [2.5 to 113.1] | 1.7 [0.5 to 5.2] | 3.0 [0.0 to 312.7] | 1.0 [1.0 to 1.0]
  anti-HPV-18, Week 10: number analyzed (Participants) | 9 | 11 | 0 | 1
  anti-HPV-18, Week 10 | 22.9 [3.4 to 152.2] | 2.3 [0.9 to 5.8] |  | 21.6 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.
  anti-HPV-18, Month 7: number analyzed (Participants) | 8 | 14 | 3 | 3
  anti-HPV-18, Month 7 | 10.1 [1.8 to 58.2] | 2.2 [1.0 to 4.8] | 44.2 [14.3 to 136.9] | 16.3 [1.0 to 265.0]
  anti-HPV-18, Month 12: number analyzed (Participants) | 9 | 15 | 2 | 1
  anti-HPV-18, Month 12 | 23.9 [8.0 to 72.0] | 2.4 [0.9 to 6.8] | 32.7 [17.2 to 62.1] | 16.3 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.
  anti-HPV-18, Month 24: number analyzed (Participants) | 7 | 10 | 3 | 1
  anti-HPV-18, Month 24 | 8.8 [1.6 to 48.5] | 1.5 [0.8 to 3.0] | 13.8 [1.3 to 149.2] | 1.0 [NA to NA] — The confidence interval could not be calculated, as there was only one participant analyzed.

33. Secondary Outcome: Frequency of Specific B-cells for HPV-16/18 Antigens
Description: B-cell memory was assessed by Enzyme Linked Immuno Spot (ELISPOT) assay. The assay was performed in a subset of approximately 100 subjects (50 HIV+ and 50 HIV-).
Time Frame: At Day 0, Week 6, Week 10, Month 7 and Month 12
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity,which included subjects in a subset of approximately 100 subjects(50 HIV+ and 50 HIV-),who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity corresponding to each time point were available.
Measure: Median (Inter-Quartile Range); unit: B-cells/million cells
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 16 | 12 | 20 | 20
B-cells/million cells
  HPV-16, Day 0: number analyzed (Participants) | 12 | 11 | 18 | 20
  HPV-16, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 61.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  HPV-18, Day 0: number analyzed (Participants) | 12 | 11 | 18 | 20
  HPV-18, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  HPV-16, Week 6: number analyzed (Participants) | 10 | 12 | 15 | 15
  HPV-16, Week 6 | 91.0 [1.0 to 154.0] | 1.0 [1.0 to 1.0] | 22.0 [1.0 to 154.0] | 1.0 [1.0 to 204.0]
  HPV-18, Week 6: number analyzed (Participants) | 10 | 12 | 15 | 15
  HPV-18, Week 6 | 39.5 [1.0 to 693.0] | 1.0 [1.0 to 45.5] | 155.0 [1.0 to 345.0] | 33.0 [1.0 to 80.0]
  HPV-16, Week 10: number analyzed (Participants) | 12 | 9 | 20 | 20
  HPV-16, Week 10 | 558.0 [95.5 to 989.5] | 198.0 [1.0 to 391.0] | 494.0 [90.5 to 834.0] | 150.5 [33.5 to 726.5]
  HPV-18, Week 10: number analyzed (Participants) | 12 | 9 | 20 | 20
  HPV-18, Week 10 | 150.0 [31.0 to 471.0] | 1.0 [1.0 to 42.0] | 211.0 [84.0 to 656.0] | 29.5 [1.0 to 222.0]
  HPV-16, Month 7: number analyzed (Participants) | 13 | 9 | 20 | 17
  HPV-16, Month 7 | 624.0 [457.0 to 1196.0] | 213.0 [165.0 to 632.0] | 1504.0 [481.0 to 3026.0] | 448.0 [257.0 to 890.0]
  HPV-18, Month 7: number analyzed (Participants) | 13 | 9 | 20 | 17
  HPV-18, Month 7 | 332.0 [153.0 to 494.0] | 1.0 [1.0 to 392.0] | 513.5 [111.5 to 1292.0] | 65.0 [1.0 to 158.0]
  HPV-16, Month 12: number analyzed (Participants) | 16 | 8 | 20 | 17
  HPV-16, Month 12 | 256.5 [75.5 to 891.5] | 121.0 [64.5 to 315.0] | 414.5 [94.5 to 640.5] | 256.0 [218.0 to 449.0]
  HPV-18, Month 12: number analyzed (Participants) | 16 | 8 | 20 | 17
  HPV-18, Month 12 | 101.0 [1.0 to 525.0] | 1.0 [1.0 to 159.0] | 250.5 [1.0 to 481.5] | 58.0 [1.0 to 101.0]

34. Secondary Outcome: Frequency of Cluster of Differentiation 4/8 [CD4+/CD8+] T-cell Response
Description: The combinations of cytokines expressed were CD4/8-all doubles, CD4/8-d-cluster of differentiation 40 Ligand (CD40L), CD4/8-d-interferon gamma (IFNG), CD4/8-interleukin-2 (IL-2), CD4/8-d-tumour necrosis alpha (TNFA), as assessed by Intracellular cytokine staining (ICS). The assay was performed in a subset of approximately 100 subjects (50 HIV+ and 50 HIV-).
Time Frame: At Day 0, Week 6, Week 10, Month 7 and Month 12
Population: The analysis was performed on the Adapted ATP cohort for immunogenicity,which included subjects in a subset of approximately 100 subjects(50 HIV+ and 50 HIV-) who met all eligibility criteria and for whom data concerning immunogenicity endpoint measures obtained from the ATP cohort for immunogenicity corresponding to each time point were available.
Measure: Median (Inter-Quartile Range); unit: CD4 cells/million T-cells
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
Number analyzed (Participants) | 17 | 15 | 21 | 19
CD4 cells/million T-cells
  CD4-All doubles,Anti-HPV-16,Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-All doubles,Anti-HPV-16,Day 0 | 41.0 [1.0 to 118.0] | 101.0 [43.0 to 215.0] | 1.0 [1.0 to 28.0] | 54.5 [1.0 to 88.0]
  CD4-All doubles,Anti-HPV-18,Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-All doubles,Anti-HPV-18,Day 0 | 7.0 [1.0 to 116.0] | 87.0 [18.0 to 184.0] | 1.0 [1.0 to 82.0] | 1.0 [1.0 to 98.0]
  CD4-All doubles,Anti-HPV-16,Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-All doubles,Anti-HPV-16,Week 6 | 445.5 [262.0 to 1028.0] | 345.5 [227.0 to 1034.0] | 298.0 [173.0 to 540.5] | 661.0 [234.0 to 982.0]
  CD4-All doubles,Anti-HPV-18,Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-All doubles,Anti-HPV-18,Week 6 | 396.0 [163.0 to 832.0] | 309.5 [203.0 to 852.0] | 237.0 [81.0 to 421.5] | 320.5 [117.0 to 524.0]
  CD4-All doubles,Anti-HPV-16,Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-All doubles,Anti-HPV-16,Week 10 | 2955.5 [1075.0 to 5200.0] | 1449.0 [922.0 to 1778.0] | 1767.0 [916.0 to 4428.0] | 1268.5 [648.0 to 2453.0]
  CD4-All doubles,Anti-HPV-18,Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-All doubles,Anti-HPV-18,Week 10 | 2036.5 [951.0 to 3123.0] | 602.0 [498.0 to 2079.0] | 1243.0 [587.0 to 3400.0] | 515.5 [414.0 to 1178.0]
  CD4-All doubles,Anti-HPV-16,Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-All doubles,Anti-HPV-16,Month 7 | 3693.0 [1870.0 to 5153.0] | 1679.5 [1052.0 to 2734.0] | 3414.5 [1424.5 to 4520.0] | 1505.0 [995.0 to 2205.0]
  CD4-All doubles,Anti-HPV-18,Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-All doubles,Anti-HPV-18,Month 7 | 1866.0 [1267.0 to 2875.0] | 840.5 [518.0 to 1641.0] | 2084.5 [911.0 to 4110.0] | 669.0 [470.0 to 1035.0]
  CD4-All doubles, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-All doubles, Anti-HPV-16, Month 12 | 2328.0 [1225.0 to 4614.0] | 1288.0 [976.0 to 2485.0] | 2543.0 [1232.0 to 4264.0] | 830.0 [367.0 to 1386.0]
  CD4-All doubles, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-All doubles, Anti-HPV-18, Month 12 | 1654.0 [836.0 to 2634.0] | 808.5 [295.0 to 1932.0] | 1641.0 [985.0 to 2939.0] | 428.0 [162.0 to 938.0]
  CD4-d-CD40L, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-CD40L, Anti-HPV-16, Day 0 | 22.0 [1.0 to 118.0] | 99.0 [60.0 to 215.0] | 1.0 [1.0 to 58.0] | 46.0 [1.0 to 81.0]
  CD4-d-CD40L, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-CD40L, Anti-HPV-18, Day 0 | 36.0 [1.0 to 81.0] | 89.0 [1.0 to 176.0] | 1.0 [1.0 to 54.0] | 13.5 [1.0 to 100.0]
  CD4-d-CD40L, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-CD40L, Anti-HPV-16, Week 6 | 426.0 [258.5 to 999.5] | 326.5 [196.0 to 1034.0] | 298.0 [209.5 to 540.0] | 582.0 [223.0 to 967.0]
  CD4-d-CD40L, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-CD40L, Anti-HPV-18, Week 6 | 403.5 [144.0 to 835.0] | 296.0 [216.0 to 840.0] | 242.5 [36.5 to 393.0] | 310.0 [95.0 to 521.0]
  CD4-d-CD40L, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-CD40L, Anti-HPV-16, Week 10 | 2893.5 [988.0 to 5006.0] | 1440.0 [882.0 to 1814.0] | 1678.0 [917.0 to 4306.0] | 1239.0 [562.0 to 2362.0]
  CD4-d-CD40L, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-CD40L, Anti-HPV-18, Week 10 | 2015.0 [944.0 to 3021.0] | 564.5 [507.0 to 2045.0] | 1051.0 [631.0 to 3317.0] | 474.5 [385.0 to 811.0]
  CD4-d-CD40L, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-CD40L, Anti-HPV-16, Month 7 | 3658.0 [1804.0 to 5070.0] | 1619.5 [1071.0 to 2600.0] | 3290.0 [1464.5 to 4387.5] | 1389.0 [949.0 to 2133.0]
  CD4-d-CD40L, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-CD40L, Anti-HPV-18, Month 7 | 1839.0 [1066.0 to 2893.0] | 833.5 [518.0 to 1605.0] | 2014.0 [979.0 to 3878.5] | 647.0 [442.0 to 981.0]
  CD4-d-CD40L, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-CD40L, Anti-HPV-16, Month 12 | 2266.0 [1178.0 to 4558.0] | 1278.0 [955.0 to 2478.0] | 2519.0 [1232.0 to 4190.0] | 862.0 [353.0 to 1197.0]
  CD4-d-CD40L, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-CD40L, Anti-HPV-18, Month 12 | 1668.0 [807.0 to 2427.0] | 808.5 [295.0 to 1914.0] | 1641.0 [984.0 to 2767.0] | 394.0 [155.0 to 913.0]
  CD4-d-IFNG, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-IFNG, Anti-HPV-16, Day 0 | 27.0 [1.0 to 63.0] | 30.0 [1.0 to 51.0] | 1.0 [1.0 to 45.0] | 39.0 [1.0 to 61.0]
  CD4-d-IFNG, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-IFNG, Anti-HPV-18, Day 0 | 4.0 [1.0 to 42.0] | 51.0 [1.0 to 59.0] | 1.0 [1.0 to 54.0] | 21.0 [1.0 to 46.0]
  CD4-d-IFNG, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-IFNG, Anti-HPV-16, Week 6 | 222.5 [117.0 to 393.0] | 116.0 [75.0 to 222.0] | 42.5 [1.0 to 127.5] | 241.5 [71.0 to 404.0]
  CD4-d-IFNG, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-IFNG, Anti-HPV-18, Week 6 | 98.0 [25.0 to 361.0] | 104.5 [35.0 to 211.0] | 1.0 [1.0 to 44.0] | 129.5 [1.0 to 182.0]
  CD4-d-IFNG, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-IFNG, Anti-HPV-16, Week 10 | 1220.0 [554.0 to 1478.0] | 450.0 [245.0 to 527.0] | 332.0 [282.0 to 1251.0] | 442.0 [160.0 to 935.0]
  CD4-d-IFNG, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-IFNG, Anti-HPV-18, Week 10 | 694.0 [342.0 to 1207.0] | 326.5 [121.0 to 455.0] | 222.0 [124.0 to 569.0] | 202.0 [122.0 to 279.0]
  CD4-d-IFNG, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-IFNG, Anti-HPV-16, Month 7 | 1513.0 [891.0 to 1993.0] | 585.5 [190.0 to 846.0] | 731.0 [267.5 to 1245.0] | 495.0 [319.0 to 859.0]
  CD4-d-IFNG, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-IFNG, Anti-HPV-18, Month 7 | 694.0 [409.0 to 868.0] | 306.0 [171.0 to 382.0] | 414.5 [245.5 to 616.5] | 198.0 [126.0 to 435.0]
  CD4-d-IFNG, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-IFNG, Anti-HPV-16, Month 12 | 452.0 [368.0 to 1097.0] | 432.0 [202.0 to 835.0] | 621.0 [239.0 to 1042.0] | 302.0 [129.0 to 555.0]
  CD4-d-IFNG, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-IFNG, Anti-HPV-18, Month 12 | 402.0 [191.0 to 585.0] | 253.5 [92.0 to 415.0] | 273.0 [88.0 to 406.0] | 98.0 [1.0 to 154.0]
  CD4-d-IL-2, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-IL-2, Anti-HPV-16, Day 0 | 43.0 [1.0 to 81.0] | 30.0 [7.0 to 121.0] | 1.0 [1.0 to 58.0] | 1.0 [1.0 to 21.0]
  CD4-d-IL-2, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-IL-2, Anti-HPV-18, Day 0 | 46.0 [1.0 to 115.0] | 37.0 [1.0 to 102.0] | 1.0 [1.0 to 31.0] | 13.5 [1.0 to 57.0]
  CD4-d-IL-2, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-IL-2, Anti-HPV-16, Week 6 | 361.0 [235.5 to 966.0] | 300.0 [234.0 to 827.0] | 245.5 [137.0 to 468.0] | 454.5 [228.0 to 816.0]
  CD4-d-IL-2, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-IL-2, Anti-HPV-18, Week 6 | 364.5 [161.0 to 858.0] | 193.5 [94.0 to 687.0] | 227.5 [131.5 to 379.5] | 286.0 [129.0 to 413.0]
  CD4-d-IL-2, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-IL-2, Anti-HPV-16, Week 10 | 2503.0 [938.0 to 4606.0] | 1221.0 [678.0 to 1584.0] | 1542.0 [776.0 to 3499.0] | 929.5 [435.0 to 2128.0]
  CD4-d-IL-2, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-IL-2, Anti-HPV-18, Week 10 | 1668.5 [635.0 to 2183.0] | 555.5 [349.0 to 1687.0] | 1183.0 [456.0 to 2311.0] | 411.0 [245.0 to 891.0]
  CD4-d-IL-2, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-IL-2, Anti-HPV-16, Month 7 | 2847.0 [1557.0 to 4064.0] | 1318.5 [672.0 to 2141.0] | 2608.5 [1147.5 to 3875.0] | 1128.0 [697.0 to 1574.0]
  CD4-d-IL-2, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-IL-2, Anti-HPV-18, Month 7 | 1522.0 [914.0 to 2285.0] | 615.0 [472.0 to 1234.0] | 1442.0 [811.0 to 3471.0] | 537.0 [341.0 to 643.0]
  CD4-d-IL-2, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-IL-2, Anti-HPV-16, Month 12 | 1792.0 [1076.0 to 4087.0] | 1040.5 [804.0 to 1972.0] | 1861.0 [1861.0 to 3754.0] | 723.0 [330.0 to 1255.0]
  CD4-d-IL-2, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-IL-2, Anti-HPV-18, Month 12 | 1170.0 [683.0 to 2375.0] | 601.5 [230.0 to 1568.0] | 1342.0 [825.0 to 2794.0] | 337.0 [243.0 to 636.0]
  CD4-d-TNFA, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-TNFA, Anti-HPV-16, Day 0 | 1.0 [1.0 to 58.0] | 71.0 [1.0 to 252.0] | 32.0 [1.0 to 74.0] | 34.0 [1.0 to 76.0]
  CD4-d-TNFA, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD4-d-TNFA, Anti-HPV-18, Day 0 | 1.0 [1.0 to 52.0] | 35.0 [1.0 to 131.0] | 25.0 [1.0 to 39.0] | 15.5 [1.0 to 83.0]
  CD4-d-TNFA, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-TNFA, Anti-HPV-16, Week 6 | 326.5 [49.5 to 714.0] | 171.0 [133.0 to 701.0] | 237.0 [89.5 to 325.0] | 337.5 [183.0 to 648.0]
  CD4-d-TNFA, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD4-d-TNFA, Anti-HPV-18, Week 6 | 234.0 [66.0 to 579.0] | 204.0 [94.0 to 539.0] | 162.5 [75.5 to 247.0] | 156.5 [72.0 to 398.0]
  CD4-d-TNFA, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-TNFA, Anti-HPV-16, Week 10 | 2086.0 [519.0 to 4016.0] | 903.5 [606.0 to 1355.0] | 1260.0 [764.0 to 3094.0] | 865.5 [453.0 to 2100.0]
  CD4-d-TNFA, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD4-d-TNFA, Anti-HPV-18, Week 10 | 1493.5 [592.0 to 2341.0] | 443.0 [248.0 to 1432.0] | 899.0 [415.0 to 2310.0] | 334.5 [203.0 to 958.0]
  CD4-d-TNFA, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-TNFA, Anti-HPV-16, Month 7 | 2688.0 [1399.0 to 3994.0] | 1109.0 [670.0 to 2066.0] | 2621.0 [1062.0 to 3652.5] | 1215.0 [792.0 to 1665.0]
  CD4-d-TNFA, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD4-d-TNFA, Anti-HPV-18, Month 7 | 1366.0 [1126.0 to 2449.0] | 598.0 [362.0 to 1522.0] | 1614.0 [760.5 to 3463.5] | 505.0 [330.0 to 683.0]
  CD4-d-TNFA, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-TNFA, Anti-HPV-16, Month 12 | 1937.0 [883.0 to 3961.0] | 1011.5 [681.0 to 2066.0] | 2344.0 [1053.0 to 3741.0] | 646.0 [344.0 to 1219.0]
  CD4-d-TNFA, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD4-d-TNFA, Anti-HPV-18, Month 12 | 1264.0 [707.0 to 2500.0] | 527.0 [174.0 to 1684.0] | 1480.0 [703.0 to 2619.0] | 358.0 [186.0 to 617.0]
  CD8-All doubles,Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-All doubles,Anti-HPV-16, Day 0 | 1.0 [1.0 to 40.0] | 1.0 [1.0 to 43.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 29.0]
  CD8-All doubles,Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-All doubles,Anti-HPV-18, Day 0 | 6.0 [1.0 to 50.0] | 23.0 [1.0 to 60.0] | 21.0 [1.0 to 54.0] | 1.0 [1.0 to 35.0]
  CD8-All doubles,Anti-HPV-16,Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-All doubles,Anti-HPV-16,Week 6 | 2.0 [1.0 to 34.5] | 13.0 [1.0 to 70.0] | 1.0 [1.0 to 14.5] | 1.0 [1.0 to 3.0]
  CD8-All doubles,Anti-HPV-18,Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-All doubles,Anti-HPV-18,Week 6 | 37.5 [9.0 to 66.5] | 2.0 [1.0 to 42.0] | 1.0 [1.0 to 42.5] | 30.5 [1.0 to 74.0]
  CD8-All doubles,Anti-HPV-16,Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-All doubles,Anti-HPV-16,Week 10 | 41.0 [1.0 to 75.0] | 3.5 [1.0 to 36.0] | 1.0 [1.0 to 54.0] | 1.0 [1.0 to 29.0]
  CD8-All doubles,Anti-HPV-18,Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-All doubles,Anti-HPV-18,Week 10 | 11.0 [1.0 to 60.0] | 1.0 [1.0 to 60.0] | 5.0 [1.0 to 84.0] | 1.0 [1.0 to 41.0]
  CD8-All doubles,Anti-HPV-16,Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-All doubles,Anti-HPV-16,Month 7 | 51.0 [18.0 to 69.0] | 9.5 [1.0 to 33.0] | 1.0 [1.0 to 74.5] | 2.0 [1.0 to 54.0]
  CD8-All doubles,Anti-HPV-18,Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-All doubles,Anti-HPV-18,Month 7 | 41.0 [1.0 to 159.0] | 30.0 [3.0 to 49.0] | 15.5 [1.0 to 106.5] | 24.0 [1.0 to 54.0]
  CD8-All doubles,Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-All doubles,Anti-HPV-16, Month 12 | 1.0 [1.0 to 23.0] | 34.0 [1.0 to 79.0] | 23.0 [1.0 to 49.0] | 1.0 [1.0 to 24.0]
  CD8-All doubles,Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-All doubles,Anti-HPV-18, Month 12 | 25.0 [1.0 to 92.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 24.0]
  CD8-d-CD40L, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-CD40L, Anti-HPV-16, Day 0 | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 7.0]
  CD8-d-CD40L, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-CD40L, Anti-HPV-18, Day 0 | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 33.0] | 1.0 [1.0 to 16.0]
  CD8-d-CD40L, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-CD40L, Anti-HPV-16, Week 6 | 1.0 [1.0 to 24.5] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0]
  CD8-d-CD40L, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-CD40L, Anti-HPV-18, Week 6 | 9.5 [1.0 to 27.5] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 36.0]
  CD8-d-CD40L, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-CD40L, Anti-HPV-16, Week 10 | 18.5 [1.0 to 73.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 41.0] | 1.0 [1.0 to 27.0]
  CD8-d-CD40L, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-CD40L, Anti-HPV-18, Week 10 | 10.5 [1.0 to 34.0] | 2.5 [1.0 to 34.0] | 26.0 [1.0 to 72.0] | 1.0 [1.0 to 30.0]
  CD8-d-CD40L, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-CD40L, Anti-HPV-16, Month 7 | 26.0 [1.0 to 63.0] | 3.0 [1.0 to 20.0] | 2.0 [1.0 to 52.0] | 1.0 [1.0 to 36.0]
  CD8-d-CD40L, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-CD40L, Anti-HPV-18, Month 7 | 4.0 [1.0 to 42.0] | 15.0 [1.0 to 31.0] | 38.0 [1.0 to 92.0] | 4.0 [1.0 to 33.0]
  CD8-d-CD40L, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-CD40L, Anti-HPV-16, Month 12 | 1.0 [1.0 to 73.0] | 31.0 [7.0 to 39.0] | 3.0 [1.0 to 30.0] | 1.0 [1.0 to 24.0]
  CD8-d-CD40L, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-CD40L, Anti-HPV-18, Month 12 | 23.0 [1.0 to 59.0] | 1.0 [1.0 to 8.0] | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 24.0]
  CD8-d-IFNG, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-IFNG, Anti-HPV-16, Day 0 | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 43.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 2.0]
  CD8-d-IFNG, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-IFNG, Anti-HPV-18, Day 0 | 6.0 [1.0 to 33.0] | 19.0 [1.0 to 47.0] | 21.0 [1.0 to 54.0] | 4.0 [1.0 to 35.0]
  CD8-d-IFNG, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-IFNG, Anti-HPV-16, Week 6 | 2.5 [1.0 to 39.5] | 17.5 [1.0 to 78.0] | 1.0 [1.0 to 14.5] | 1.0 [1.0 to 11.0]
  CD8-d-IFNG, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-IFNG, Anti-HPV-18, Week 6 | 27.5 [1.0 to 55.5] | 1.0 [1.0 to 47.0] | 1.0 [1.0 to 42.5] | 35.5 [1.0 to 84.0]
  CD8-d-IFNG, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-IFNG, Anti-HPV-16, Week 10 | 34.0 [1.0 to 99.0] | 25.0 [1.0 to 30.0] | 1.0 [1.0 to 38.0] | 1.0 [1.0 to 29.0]
  CD8-d-IFNG, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-IFNG, Anti-HPV-18, Week 10 | 3.0 [1.0 to 68.0] | 7.5 [1.0 to 34.0] | 24.0 [1.0 to 76.0] | 1.0 [1.0 to 1.0]
  CD8-d-IFNG, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-IFNG, Anti-HPV-16, Month 7 | 46.0 [1.0 to 68.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 74.5] | 1.0 [1.0 to 50.0]
  CD8-d-IFNG, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-IFNG, Anti-HPV-18, Month 7 | 41.0 [1.0 to 68.0] | 21.0 [1.0 to 41.0] | 4.0 [1.0 to 90.5] | 3.0 [1.0 to 52.0]
  CD8-d-IFNG, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-IFNG, Anti-HPV-16, Month 12 | 1.0 [1.0 to 31.0] | 25.0 [1.0 to 57.0] | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 24.0]
  CD8-d-IFNG, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-IFNG, Anti-HPV-18, Month 12 | 23.0 [1.0 to 92.0] | 1.0 [1.0 to 31.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 4.0]
  CD8-d-IL-2, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-IL-2, Anti-HPV-16, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.0]
  CD8-d-IL-2, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-IL-2, Anti-HPV-18, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-IL-2, Anti-HPV-16, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-IL-2, Anti-HPV-18, Week 6 | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-IL-2, Anti-HPV-16, Week 10 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-IL-2, Anti-HPV-18, Week 10 | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-IL-2, Anti-HPV-16, Month 7 | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 37.5] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-IL-2, Anti-HPV-18, Month 7 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-IL-2, Anti-HPV-16, Month 12 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8-d-IL-2, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-IL-2, Anti-HPV-18, Month 12 | 1.0 [1.0 to 48.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 1.0]
  CD8-d-TNFA, Anti-HPV-16, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-TNFA, Anti-HPV-16, Day 0 | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 29.0]
  CD8-d-TNFA, Anti-HPV-18, Day 0: number analyzed (Participants) | 17 | 15 | 17 | 18
  CD8-d-TNFA, Anti-HPV-18, Day 0 | 6.0 [1.0 to 50.0] | 7.0 [1.0 to 54.0] | 1.0 [1.0 to 33.0] | 1.0 [1.0 to 34.0]
  CD8-d-TNFA, Anti-HPV-16, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-TNFA, Anti-HPV-16, Week 6 | 1.0 [1.0 to 46.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 31.0]
  CD8-d-TNFA, Anti-HPV-18, Week 6: number analyzed (Participants) | 16 | 14 | 16 | 18
  CD8-d-TNFA, Anti-HPV-18, Week 6 | 19.0 [1.0 to 50.0] | 1.0 [1.0 to 57.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 26.0]
  CD8-d-TNFA, Anti-HPV-16, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-TNFA, Anti-HPV-16, Week 10 | 1.5 [1.0 to 32.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 31.0] | 1.0 [1.0 to 26.0]
  CD8-d-TNFA, Anti-HPV-18, Week 10: number analyzed (Participants) | 14 | 14 | 19 | 18
  CD8-d-TNFA, Anti-HPV-18, Week 10 | 17.5 [1.0 to 34.0] | 14.0 [1.0 to 61.0] | 5.0 [1.0 to 42.0] | 1.0 [1.0 to 34.0]
  CD8-d-TNFA, Anti-HPV-16, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-TNFA, Anti-HPV-16, Month 7 | 34.0 [1.0 to 41.0] | 13.0 [1.0 to 33.0] | 1.0 [1.0 to 49.0] | 2.0 [1.0 to 33.0]
  CD8-d-TNFA, Anti-HPV-18, Month 7: number analyzed (Participants) | 13 | 14 | 16 | 17
  CD8-d-TNFA, Anti-HPV-18, Month 7 | 41.0 [1.0 to 111.0] | 26.5 [15.0 to 58.0] | 1.0 [1.0 to 58.0] | 1.0 [1.0 to 32.0]
  CD8-d-TNFA, Anti-HPV-16, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-TNFA, Anti-HPV-16, Month 12 | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 54.0] | 28.0 [1.0 to 49.0] | 1.0 [1.0 to 42.0]
  CD8-d-TNFA, Anti-HPV-18, Month 12: number analyzed (Participants) | 15 | 14 | 21 | 19
  CD8-d-TNFA, Anti-HPV-18, Month 12 | 30.0 [24.0 to 62.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 48.0] | 1.0 [1.0 to 40.0]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: During the 7-day follow-up period (from the day of vaccination up to 6 subsequent days) after vaccination; Unsolicited AEs: During the 30-day follow-up period (from the day of vaccination up to 29 subsequent days) after vaccination; SAEs: during the whole study period (from Day 0 up to Month 24).
Arm/Group | HIV+/Cervarix Group | HIV+/Gardasil Group | HIV-/Cervarix Group | HIV-/Gardasil Group
All-Cause Mortality (participants affected / at risk) | 0/129 | 1/128 | 0/144 | 0/145
Serious Adverse Events (participants affected / at risk) | 9/129 | 9/128 | 4/144 | 1/145
Other Adverse Events (participants affected / at risk) | 123/129 | 109/128 | 136/144 | 127/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+/Cervarix Group (N=129) | HIV+/Gardasil Group (N=128) | HIV-/Cervarix Group (N=144) | HIV-/Gardasil Group (N=145)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginitis gardnerella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+/Cervarix Group (N=129) | HIV+/Gardasil Group (N=128) | HIV-/Cervarix Group (N=144) | HIV-/Gardasil Group (N=145)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (64) | 38 (56) | 31 (40) | 34 (47)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cd4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervicitis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 4 (5) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 41 (59) | 34 (50) | 52 (89) | 42 (69)
Fatigue (General disorders) | 73 (128) | 59 (118) | 65 (111) | 56 (88)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 41 (58) | 35 (55) | 28 (35) | 26 (38)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 88 (165) | 63 (116) | 70 (115) | 67 (104)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 68 (115) | 51 (81) | 64 (106) | 54 (91)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4) | 4 (5) | 2 (3) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 121 (303) | 85 (174) | 133 (329) | 119 (265)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 24 (32) | 20 (22) | 23 (31) | 25 (29)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 5 (6) | 5 (6) | 8 (10)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 38 (60) | 21 (28) | 47 (76) | 39 (60)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 4 (5)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 14 (17) | 9 (11) | 4 (6) | 6 (7)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral load increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.